CLINICAL TRIAL: NCT02020889
Title: A Double-blind, Randomised, Placebo-controlled Study to Investigate the Efficacy and Safety of Mepolizumab in the Treatment of Eosinophilic Granulomatosis With Polyangiitis in Subjects Receiving Standard of Care Therapy
Brief Title: A Study to Investigate Mepolizumab in the Treatment of Eosinophilic Granulomatosis With Polyangiitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115921
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Churg-Strauss Syndrome
Keywords: eosinophils; SB 240563; Churg-Strauss Syndrome; quality of life; mepolizumab; safety; biomarkers; efficacy; corticosteroids; Eosinophilic granulomatosis with polyangiitis
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mepolizumab 300 mg (Experimental): Each subject will receive mepolizumab 300 mg subcutaneous (SC) injection every 4 weeks (13 administrations) along with standard care. It will be administered as 3 separate injections (100 mg each- total dose 300 mg); individual injection sites will be separated by at least 5 cm. It will be administered into any of the upper arm, thigh or anterior abdominal wall.
  Interventions: Biological: Mepolizumab
- Placebo (Placebo Comparator): Each subject will receive placebo (0.9% sodium chloride) SC injection every 4 weeks (13 administrations) along with standard care. It will be administered as 3 separate injections; individual injection sites will be separated by at least 5 cm. It will be administered into any of the upper arm, thigh or anterior abdominal wall.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab will be provided as a lyophilized cake in sterile vials for individual use to be reconstituted with sterile water for Injection, just prior to use.
  Arms: Mepolizumab 300 mg
Drug: Placebo — Placebo will be available as 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double-blind study is to investigate the efficacy and safety of mepolizumab (300 milligram [mg] administered subcutaneously [SC] every 4 weeks) compared with placebo over a 52-week study treatment period in subjects with relapsing or refractory Eosinophilic Granulomatosis with Polyangiitis (EGPA) receiving standard of care therapy including background corticosteroid therapy with or without immunosuppressive therapy. During the treatment period, in accordance with standard of care, corticosteroid dose will be tapered. The key outcomes in the study focus on evaluation of clinical remission, defined as Birmingham Vasculitis Activity Score (BVAS)=0 with a corticosteroid dose of <=4 mg/day prednisolone/prednisone, reduction in disease relapse and reduction in corticosteroid requirement.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Age and gender: Male or female subjects age 18 years or older.
* EGPA diagnosis: subjects who have been diagnosed with EGPA for at least 6 months based on the history or presence of: asthma plus eosinophilia (>1.0x10^9/Liter and/or >10% of leucocytes) plus at least two of the following additional features of EGPA; a biopsy showing histopathological evidence of eosinophilic vasculitis, or perivascular eosinophilic infiltration, or eosinophil-rich granulomatous inflammation; neuropathy, mono or poly (motor deficit or nerve conduction abnormality); pulmonary infiltrates, non-fixed; sino-nasal abnormality; cardiomyopathy (established by echocardiography or Magnetic Resonance Imaging); glomerulonephritis (haematuria, red cell casts, proteinuria); alveolar haemorrhage (by bronchoalveolar lavage); palpable purpura; anti neutrophil cytoplasmic anti-body (ANCA) positive (Myeloperoxidase or proteinease 3).
* History of relapsing OR refractory disease defined as: Relapsing disease:

Subject must have a past history of at least one confirmed EGPA relapse (i.e., requiring increase in oral corticosteroids (OCS) dose, initiation/increased dose of immunosuppressive therapy or hospitalisation) within the past 2 years which occurred at least 12 weeks prior to Screening (Visit 1) whilst receiving a dose of prednisolone (or equivalent) of >=7.5 milligram per day (mg/day). Refractory disease: Either: Failure to attain remission (BVAS=0 and OCS dose <=7.5 mg/day prednisolone or equivalent) within the last 6 months following induction treatment with a standard regimen, administered for at least 3 months. Note: a) Subjects who have received a cyclophosphamide (CYC) induction regimen may be included a minimum of 2 weeks after the last dose of daily oral CYC, or 3 weeks after the last dose of pulsed intravenous CYC prior to Baseline (Visit 2), if their total white blood cells (WBC) is >=4x10^9/Liter (tested at the local laboratory, if necessary) prior to randomisation. b) Subjects who have received a methotrexate, azathioprine, or mycophenolate mofetil induction regimen may be included if on a stable dose for at least 4 weeks prior to Baseline (Visit 2). c) Subjects who have received an induction regimen comprising corticosteroids alone may be included only if they have failed to attain remission after 3 months of treatment AND the corticosteroid dose is >=15 mg/day prednisolone or equivalent for the 4 weeks prior to Baseline (Visit 2). Or: Within 6 months prior to Screening (Visit 1), recurrence of symptoms of EGPA (not necessarily meeting the protocol definition of relapse) whilst tapering OCS, occurring at any dose level >=7.5 mg/day prednisolone or equivalent.

* Corticosteroid therapy: Subject must be on a stable dose of oral prednisolone or prednisone of >=7.5 mg/day (but not >50 mg/day) for at least 4 weeks prior to Baseline (Visit 2).
* Immunosuppressive therapy: If receiving immunosuppressive therapy (excluding cyclophosphamide) the dosage must be stable for the 4 weeks prior to Baseline (Visit 2) and during the study (dose reductions for safety reasons will be permitted).
* ECG measurements: QTc(F)<450 msec or QTc(F)<480 msec for patients with bundle branch block. The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual overread. For subject eligibility and withdrawal decisions, QTcFwill be used. For purposes of data analysis, QTcF will be used as primary though data using both correction formulas will be collected and analysed. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.
* Female subjects: To be eligible for entry into the study, females of childbearing potential (FCBP) must commit to consistent and correct use of an acceptable method of birth control (as discussed in the protocol) beginning with consent, for the duration of the trial and for 4 months after the last study drug administration.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* Liver Function Tests: obtained at Screening (Visit 1): ALT<2x ULN (upper limit of normal) or if subject is on background methotrexate or azathioprine <3x ULN; AST<2x ULN or if subject is on background methotrexate or azathioprine <3x ULN; Alkaline Phosphatase ≤2.0x ULN;Bilirubin ≤ 1.5x ULN (isolated bilirubin>1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)

Exclusion Criteria:

* GPA or MPA: Diagnosed with granulomatosis with polyangiitis (GPA; previously known as Wegener's granulomatosis) or microscopic polyangiitis (MPA).
* Organ-threatening EGPA: Organ-threatening EGPA as per European league against rheumatism (EULAR) criteria, i.e., organ failure due to active vasculitis, creatinine >5.8 gram per deciliter (g/dL) (>513 micromole per liter [µmol/L]) within 3 months prior to Screening (Visit 1).
* Life-threatening EGPA: Imminently life-threatening EGPA disease defined as any of the following within 3 months prior to Screening (Visit 1); Intensive care required; Severe alveolar haemorrhage or haemoptysis requiring transfusion or ventilation or haemoglobin < 8 gram per liter (g/dL) (<80 g/L) or drop in haemoglobin > 2 g/dL (>20 g/L) over a 48 hour period due to alveolar haemorrhage; Rapidly progressive glomerulonephritis (RPGN) with creatinine > 2.5 milligram per deciliter (mg/dL) (>221 µmol/L) or rise in creatinine > 2 mg/dL (>177 µmol/L) over a 48 hour period; Severe gastrointestinal (GI) involvement, e.g., gangrene, bleeding requiring surgery; Severe central nervous system (CNS) involvement; Severe cardiac involvement, e.g., life-threatening arrhythmia, cardiac failure: ejection fraction < 20%, New York Heart Association Class III/IV (as discussed in protocol), acute myocardial infarction.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior screening (Subjects that had localized carcinoma (i.e., basal or squamous cell) of the skin which was resected for cure will not be excluded).
* Liver disease: Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, and known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Cardiovascular: Subjects who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment including but not limited to: Known ejection fraction of <30%, OR Severe heart failure that meets New York Heart Association Class IV (as discussed in protocol), OR Hospitalised in the 12 months prior to Visit 1 for severe heart failure meeting New York Heart Association Class III (as discussed in protocol), OR Angina diagnosed less than 3 months prior to or at Visit 1 (Screening).
* Other concurrent medical conditions: Subjects who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological, respiratory or any other system abnormalities that are not associated with EGPA and are uncontrolled with standard treatment.
* Infectious disease: Chronic or ongoing active infectious disease requiring systemic treatment.
* Parasitic infection: Subjects with a parasitic infestation within 6 months prior to Screening (Visit 1).
* Hepatitis status: Diagnosis of chronic hepatitis B, as evidenced by positive Hepatitis B surface antigen (HBsAg) at Screening (Visit 1). Japan only: Subjects positive for HBsAg , antibodies to HBsAg, i.e., HBsAb, or Hepatitis B core antigen, i.e., HBcAb, at Screening (Visit 1). Note: Subjects with antibodies to HBsAg, i.e., HBsAb positive, only (i.e., negative for HBsAg and HBcAb) with a history of hepatitis B vaccination can be included.
* HIV: Subjects with a known human immunodeficiency virus infection.
* Hypersensitivity: Subjects with a known allergy or intolerance to a monoclonal antibody or biologic therapy.
* Previous mepolizumab: Subjects who have previously received mepolizumab within a 1 year period prior to Screening (Visit 1).
* Prohibited medications: Subjects receiving any of the following: OCS: Subject requires an oral corticosteroid dose of >50 mg/day prednisolone/prednisone in the 4-week period prior to Baseline (Visit 2); Intravenous or SC corticosteroids in the 4-week period prior to Baseline (Visit 2); Omalizumab within 130 days prior to Screening (Visit 1); Cyclophosphamide: oral CYC within 2 weeks prior to Baseline (Visit 2) and IV CYC within 3 weeks prior to Baseline (Visit 2), if their total WBC is >=4x10^9/Liter (measured using the local laboratory if necessary); Rituximab within 12 months prior to Screening (Visit 1); in addition, the subject must have shown recovery of peripheral B-cell count to within the normal range; IV or SC immunoglobulin within 6 months prior to Screening (Visit 1); Interferon-α within 6 months prior to Screening (Visit 1); Anti-TNF therapy within 12 weeks prior to Screening (Visit 1); Anti-CD52 (alemtuzumab) within 6 months prior to Screening (Visit 1).
* Other laboratory parameter exclusions: Creatinine > 2.5 mg/dL (221 µmol/L); WBC < 4 x10^9/Liter, Platelet count <120,000/millimetre cube (mm^3), Haemoglobin <8 g/dL (<80 g/L)
* Pregnancy: Subjects who are pregnant or breastfeeding. Subjects should not be enrolled if they plan to become pregnant during the time of study participation.
* Alcohol/substance abuse: A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Screening (Visit 1).
* Other investigational product: Subjects who have received treatment with an investigational drug within the past 30 days or 5 terminal phase half-lives of the drug whichever is longer, prior to Screening (Visit 1) (this also includes investigational formulations of marketed products).
* Other clinical study: Subject is currently participating in any other interventional clinical study.
* Adherence: Subjects who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.
* French subjects: the French subject has participated in any study using an investigational drug during the previous 30 days or 5 half-lives (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2016-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (7):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Salt Lake City, Utah
- GSK Investigational Site, Brussels, Belgium
- Canada (2):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
- France (5):
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Suresnes
- Germany (6):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Kirchheim unter Teck
- Italy (3):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Pisa, Tuscany
- Japan (2):
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
- GSK Investigational Site, Barcelona, Spain
- United Kingdom (3):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, Portsmouth

REFERENCES:
- [Derived] Wechsler ME, Akuthota P, Jayne D, Khoury P, Klion A, Langford CA, Merkel PA, Moosig F, Specks U, Cid MC, Luqmani R, Brown J, Mallett S, Philipson R, Yancey SW, Steinfeld J, Weller PF, Gleich GJ; EGPA Mepolizumab Study Team. Mepolizumab or Placebo for Eosinophilic Granulomatosis with Polyangiitis. N Engl J Med. 2017 May 18;376(20):1921-1932. doi: 10.1056/NEJMoa1702079. PMID 28514601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants at screening and run-in visit, entered a 52 week study treatment phase followed by 8-week follow-up phase. The total duration for the study participation was approximately 64 weeks.
Pre-assignment Details: A total of 151 participants with a history of relapsing or refractory Eosinophilic Granulomatosis with Polyangiitis (EGPA) were screened, out of which 4 were screen failures and 11 were run-in failures. 136 participants completed run-in period and received Mepolizumab 300 milligram (mg) or placebo in a randomized manner in the treatment phase.
Groups:
- Placebo: Participants received placebo injection via subcutaneous (SC) route once every 4 weeks along with standard of care (SOC) drugs up to Week 48.
- Mepolizumab 300mg: Participants received Mepolizumab 300mg injection via SC route once every 4 weeks along with SOC drugs up to Week 48.
Period: Overall Study
Arm/Group | Placebo | Mepolizumab 300mg
Started | 68 | 68
Completed | 61 | 65
Not Completed | 7 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mepolizumab 300mg | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (14.32) | 48.7 (12.39) | 48.5 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 80
  Male | 30 | 26 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: American Indian or Alaskan Native | 0 | 1 | 1
  Race customized: Asian - Japanese Heritage | 3 | 3 | 6
  Race customized: Asian - South East Asian Heritage | 2 | 0 | 2
  Race customized: White - Arabic/North African Heritage | 0 | 2 | 2
  Race customized: White - White/Caucasian/European Heritage | 61 | 62 | 123
  Race customized: Mixed Race | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Category of Accrued Duration of Remission
Description: Total accrued duration of remission is the accrued number of weeks where Birmingham Vasculitis Activity Score (BVAS) =0 plus prednisolone/prednisone dose <=4 mg/day over the 52 week study treatment period was reported. The accrued duration was categorized into zero, >0 to <12 weeks, 12 to <24 weeks, 24 to <36 weeks and >=36 weeks. Statistical analysis was based on a proportional odds regression model with covariates including treatment group, Baseline prednisolone/prednisone daily dose, Baseline BVAS score and region. Intent-to-Treat (ITT) Population was used for the analysis and was defined as all participants who were randomized and received at least one dose of trial medication. Randomized participants were assumed to have received study treatment unless definitive evidence to the contrary exists. The odds ratio for treatment difference and associated probability (p)-value and 95 percent confidence interval (CI) were calculated.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants
  Zero | 55 | 32
  >0 to <12 weeks | 8 | 8
  12 to <24 weeks | 3 | 9
  24 to <36 weeks | 0 | 10
  >=36 weeks | 2 | 9
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p < 0.001, Proportional odds regression model; Proportional odds regression model with covariates including treatment group, Baseline prednisolone/prednisone daily dose, Baseline BVAS score, region; Odds Ratio (OR) = 5.91, 95% CI 2-sided [2.68 to 13.03] — Mepolizumab 300mg/Placebo

2. Primary Outcome: Number of Participants Who Are in Remission at 36 and 48 Weeks
Description: The number of participants who were in remission (i.e ., BVAS=0 and prednisolone /prednisone <=4 mg/day) at both Weeks 36 and 48 of the study treatment period was reported. The statistical analysis was performed using a logistic regression model on ITT Population. The odds ratio for treatment difference and associated p-value and 95 percent CI were calculated.
Time Frame: Week 36 and Week 48
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants | 2 | 22
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p < 0.001, Regression, Logistic; Logistic regression model with covariates including treatment group, Baseline prednisolone/prednisone daily dose, Baseline BVAS score and region; Odds Ratio (OR) = 16.74, 95% CI 2-sided [3.61 to 77.56] — Mepolizumab 300mg/Placebo

3. Secondary Outcome: Time to First EGPA Relapse
Description: EGPA relapse was defined as worsening or persistence of active disease since the last visit characterized by active vasculitis or active asthma symptoms and/or signs with a corresponding worsening in Asthma Control Questionnaire-6 (ACQ-6) score or active nasal and/or sinus disease, with a corresponding worsening in at least one of the sino-nasal symptom questions warranting: i) an increased dose of OCS therapy (or other systemic corticosteroid therapy) to >4 mg/day prednisolone total daily dose or equivalent; OR ii) an increased dose or addition of immunosuppressive therapy; OR iii) hospitalization related to EGPA worsening. Participants who completed study, or withdrawn prematurely from the study without experiencing the event were censored. The number of participants with at least one EGPA relapse during the planned study treatment period are presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants | 56 | 38
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p < 0.001, Cox Proportional Hazard regression; Cox proportional hazards model with covariates of treatment group, Baseline prednisolone/prednisone daily dose, Baseline BVAS score and region; Hazard Ratio (HR) = 0.322, 95% CI 2-sided [0.206 to 0.502] — Mepolizumab 300mg/Placebo

4. Secondary Outcome: Number of Participants in Each Category of Average Daily Prednisolone/Prednisone Dose During the Last 4 Weeks of the Study Treatment Period.
Description: The number of participants with an average daily prednisolone/prednisone dose during the last 4 weeks of the Study Treatment Period (48 through 52) was calculated. The average dose was categorized into zero, >0 to <=4.0mg, >4.0 to <=7.5mg and >7.5mg. The statistical analysis was performed using a proportional odds regression model with Baseline covariates of treatment group, Baseline prednisolone/prednisone daily dose, Baseline BVAS score and region and the comparison between treatment groups was presented as an odds ratio, p-value and 95 percent CI.
Time Frame: Week 48 and Week52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants
  Zero | 2 | 12
  >0 to <=4.0mg | 3 | 18
  >4.0 to <=7.5mg | 18 | 10
  >7.5mg | 45 | 28
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p < 0.001, Proportional odds regression model; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.20, 95% CI 2-sided [0.09 to 0.41] — Mepolizumab 300mg/Placebo

5. Secondary Outcome: Number of Participants Who Achieved Remission Within the First 24 Weeks and Remained in Remission for the Remainder of the Treatment Period
Description: The number of participants who achieved remission (i.e., BVAS=0 and prednisolone/prednisone<=4 mg/day) within the first 24 weeks and remain in remission for the remainder of the study treatment period was reported. The statistical analysis was performed using a logistic regression model on ITT Population. The odds ratio for treatment difference and associated p-value and 95 percent CI were calculated.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants | 1 | 13
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p = 0.007, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 19.65, 95% CI 2-sided [2.30 to 167.93] — Mepolizumab 300mg/Placebo

6. Secondary Outcome: Number of Participants in Each Category of Accrued Duration of Remission
Description: Total accrued duration of remission, i.e., the accrued number of weeks where Birmingham Vasculitis Activity Score (BVAS) =0 plus prednisolone/prednisone dose <=7.5mg/day over the 52 week study treatment period was reported. BVAS is a validated, clinician-completed tool used for the comprehensive multisystem clinical assessment of disease activity in systemic vasculitis. The duration was categorized into zero, >0 to <12 weeks, 12 to <24 weeks, 24 to <36 weeks and >=36 weeks. Statistical analysis was performed on ITT Population and was based on a proportional odds regression model with covariates including treatment group, Baseline prednisolone/prednisone daily dose, Baseline BVAS score and region. The odds ratio for treatment difference and associated p-value and 95 percent CI were calculated.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants
  Zero | 36 | 15
  >0 to <12 weeks | 19 | 15
  12 to <24 weeks | 0 | 7
  24 to <36 weeks | 7 | 9
  >=36 weeks | 6 | 22
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p < 0.001, Proportional odds regression model; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.31, 95% CI 2-sided [2.63 to 10.74] — Mepolizumab 300mg/Placebo

7. Secondary Outcome: Number of Participants Who Are in Remission at 36 and 48 Weeks
Description: The number of participants who were in remission (i.e ., BVAS=0 and prednisolone /prednisone <=7.5mg/day) at both Weeks 36 and 48 of the study treatment period was reported. The statistical analysis was performed using a logistic regression model on ITT Population. The odds ratio for treatment difference and associated p-value and 95 percent CI were calculated.
Time Frame: Week 36 and Week 48
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants | 7 | 28
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 7.19, 95% CI 2-sided [2.60 to 19.87] — Mepolizumab 300mg/Placebo

8. Secondary Outcome: Number of Participants Who Achieved Remission (BVAS=0 and Prednisolone/Prednisone <=7.5 mg/Day) Within the First 24 Weeks and Remained in Remission for the Remainder of the Treatment Period
Description: as for outcome 7
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants | 2 | 16
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 300mg; Test type: Other; p = 0.003, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 11.39, 95% CI 2-sided [2.35 to 55.24] — Mepolizumab 300mg/Placebo

9. Secondary Outcome: Number of Participants With Local and Systemic Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs including systemic allergic and non-allergic reactions as well as local site injection-related reactions were counted throughout treatment phase and follow up phase. Systemic allergic reactions included Facial paralysis, flushing, hypersensitivity and rash pruritic. Injection related reactions were considered as systemic non-allergic reactions. Local site reactions included injection site bruising, erythema, pain and reaction. The analysis was performed on Safety Population which comprised of all participants who receive at least one dose of study treatment.
Time Frame: Up to Week 52
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Participants
  Facial paralysis | 1 | 0
  Flushing | 0 | 1
  Hypersensitivity | 0 | 1
  Rash pruritic | 0 | 1
  Injection related reactions | 0 | 1
  Injection site bruising | 0 | 1
  Injection site erythema | 1 | 1
  Injection site pain | 1 | 0
  Injection site reaction | 7 | 9

10. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters of Alanine Aminotransferase (ALT), Alkaline Phosphatase (Alk.Phosph.), Aspartate Aminotransferase (AST), Creatinine Kinase, Gamma Glutamyl Transaminase (GGT) and Lactate Dehydrogenase (Dehydro) Levels
Description: Blood samples were collected to evaluate change from Baseline in ALT, Alk.phosph., AST, creatinine kinase, GGT and lactate dehydro values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety population
Measure: Mean (Standard Deviation); unit: International Unit per Liter (IU/L)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
International Unit per Liter (IU/L)
  Absolute ALT; Baseline; n= 68, 68 | 19.9 (8.91) | 21.3 (14.22)
  ALT; Week 4; n= 68, 68 | 0.2 (6.17) | -2.2 (8.59)
  ALT; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  ALT; Week 8; n= 67, 66 | -0.9 (5.66) | -1.7 (10.14)
  ALT; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  ALT; Week 12; n= 65, 68 | -0.9 (4.53) | -0.7 (12.65)
  ALT; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  ALT; Week 16; n= 65, 68 | -0.4 (6.56) | -2.2 (9.73)
  ALT; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  ALT; Week 20; n= 63, 68 | -0.3 (6.25) | -1.2 (12.30)
  ALT; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  ALT; Week 24; n= 63, 66 | -1.3 (5.38) | -0.2 (15.77)
  ALT; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  ALT; Week 28; n= 62, 66 | -0.9 (6.73) | -0.4 (13.62)
  ALT; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  ALT; Week 32; n= 61, 67 | -0.7 (6.79) | -2.4 (11.30)
  ALT; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  ALT; Week 36; n= 60, 67 | -0.1 (6.21) | -3.0 (11.66)
  ALT; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  ALT; Week 40; n= 61, 66 | 0.3 (9.01) | -2.3 (11.70)
  ALT; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  ALT; Week 44; n= 61, 66 | 0.9 (9.68) | -2.7 (9.51)
  ALT; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  ALT; Week 48; n= 61, 64 | 1.7 (9.04) | -1.6 (15.47)
  ALT; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  ALT; Week 52; n= 60, 65 | 1.5 (10.42) | -2.8 (12.87)
  ALT; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  ALT; Week 56; n= 61, 63 | -0.1 (7.35) | -3.6 (12.79)
  ALT; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  ALT; Week 60; n= 60, 65 | -0.3 (7.33) | -4.7 (14.11)
  Absolute Alk.phosph.; Baseline; n= 68, 68 | 61.2 (17.83) | 60.4 (20.90)
  Alk.phosph.; Week 4; n= 68, 68 | -0.9 (6.65) | -3.2 (10.01)
  Alk.phosph.; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Alk.phosph.; Week 8; n= 67, 66 | -1.7 (9.95) | -1.7 (11.56)
  Alk. phosph.; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Alk. phosph.; Week 12; n= 65, 68 | -1.9 (8.36) | -1.1 (12.99)
  Alk. phosph.; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Alk. phosph.; Week 16; n= 65, 68 | -1.3 (9.35) | -1.1 (14.61)
  Alk. phosph.; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Alk. phosph.; Week 20; n= 63, 68 | 0.0 (11.24) | 4.4 (21.90)
  Alk. phosph.; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Alk. phosph.; Week 24; n= 63, 66 | -1.1 (10.65) | 2.8 (17.64)
  Alk. phosph.; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Alk. phosph.; Week 28; n= 62, 66 | 0.2 (10.95) | 4.9 (17.17)
  Alk. phosph.; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Alk. phosph.; Week 32; n= 61, 67 | 0.2 (11.14) | 4.4 (15.83)
  Alk. phosph.; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Alk. phosph.; Week 36; n= 60, 67 | 0.2 (10.42) | 4.8 (14.71)
  Alk. phosph.; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Alk. phosph.; Week 40; n= 61, 66 | 1.0 (10.08) | 6.2 (18.43)
  Alk. phosph.; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Alk. phosph.; Week 44; n= 61, 66 | 1.1 (12.55) | 5.1 (16.53)
  Alk. phosph.; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Alk. phosph.; Week 48; n= 61, 64 | 1.2 (11.66) | 5.1 (17.56)
  Alk. phosph.; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Alk. phosph.; Week 52; n= 60, 65 | 0.3 (12.30) | 2.3 (14.47)
  Alk. phosph.; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Alk. phosph.; Week 56; n= 61, 63 | -0.9 (12.04) | 1.7 (16.42)
  Alk. phosph.; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Alk. phosph.; Week 60; n= 60, 65 | -1.5 (13.16) | 1.0 (15.08)
  Absolute AST; Baseline; n= 68, 68 | 19.3 (6.11) | 21.8 (10.73)
  AST; Week 4; n= 68, 68 | 0.0 (4.41) | -1.7 (8.61)
  AST; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  AST; Week 8; n= 67, 66 | -0.4 (4.77) | -1.0 (8.21)
  AST; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  AST; Week 12; n= 65, 68 | 0.5 (4.41) | -0.7 (9.62)
  AST; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  AST; Week 16; n= 65, 68 | 0.4 (5.48) | -0.6 (7.90)
  AST; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  AST; Week 20; n= 63, 68 | 0.8 (4.66) | -0.6 (8.49)
  AST; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  AST; Week 24; n= 63, 66 | 0.0 (4.46) | -0.4 (10.44)
  AST; Week 28; n= 61, 66: number analyzed (Participants) | 61 | 66
  AST; Week 28; n= 61, 66 | -0.9 (5.34) | -0.4 (10.59)
  AST; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  AST; Week 32; n= 61, 67 | -0.2 (4.91) | -1.3 (10.67)
  AST; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  AST; Week 36; n= 60, 67 | 0.2 (4.68) | -2.2 (9.61)
  AST; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  AST; Week 40; n= 61, 66 | 0.5 (5.51) | -1.6 (8.97)
  AST; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  AST; Week 44; n= 61, 66 | 0.4 (5.77) | -2.4 (9.02)
  AST; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  AST; Week 48; n= 61, 64 | 1.1 (6.86) | -2.3 (10.14)
  AST; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  AST; Week 52; n= 60, 65 | 0.9 (6.84) | -3.0 (10.49)
  AST; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  AST; Week 56; n= 61, 63 | -0.2 (4.92) | -2.8 (10.64)
  AST; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  AST; Week 60; n= 60, 65 | -0.4 (5.24) | -3.7 (10.92)
  Absolute Creatinine kinase; Baseline; n= 68, 68 | 99.0 (75.99) | 88.8 (75.18)
  Creatinine kinase; Week 4; n= 68, 68 | -2.4 (83.23) | 2.0 (60.92)
  Creatinine kinase; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Creatinine kinase; Week 8; n= 67, 66 | -5.0 (62.41) | 3.5 (50.48)
  Creatinine kinase; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Creatinine kinase; Week 12; n= 65, 68 | 5.4 (93.24) | 6.1 (40.86)
  Creatinine kinase; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Creatinine kinase; Week 16; n= 65, 68 | 15.8 (125.84) | 0.5 (49.65)
  Creatinine kinase; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Creatinine kinase; Week 20; n= 63, 68 | 1.3 (78.35) | 6.5 (54.83)
  Creatinine kinase; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Creatinine kinase; Week 24; n= 63, 66 | -0.6 (56.55) | 6.0 (66.69)
  Creatinine kinase; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Creatinine kinase; Week 28; n= 62, 66 | -15.9 (59.38) | 6.3 (55.84)
  Creatinine kinase; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Creatinine kinase; Week 32; n= 61, 67 | -13.1 (59.29) | 0.2 (49.68)
  Creatinine kinase; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Creatinine kinase; Week 36; n= 60, 67 | -12.0 (65.11) | 4.9 (52.71)
  Creatinine kinase; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Creatinine kinase; Week 40; n= 61, 66 | 2.6 (91.89) | 2.8 (62.74)
  Creatinine kinase; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Creatinine kinase; Week 44; n= 61, 66 | 5.8 (86.76) | -2.4 (62.13)
  Creatinine kinase; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Creatinine kinase; Week 48; n= 61, 64 | -8.1 (70.09) | -2.6 (90.09)
  Creatinine kinase; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Creatinine kinase; Week 52; n= 60, 65 | 0.9 (67.51) | 0.2 (53.45)
  Creatinine kinase; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Creatinine kinase; Week 56; n= 61, 63 | -8.7 (60.58) | -0.2 (62.08)
  Creatinine kinase; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Creatinine kinase; Week 60; n= 60, 65 | -10.3 (65.83) | 0.4 (61.45)
  Absolute GGT; Baseline; n= 68, 68 | 30.8 (25.49) | 30.1 (27.24)
  GGT; Week 4; n= 68, 68 | 0.2 (11.70) | -2.0 (9.68)
  GGT; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  GGT; Week 8; n= 67, 66 | -1.0 (8.59) | -0.6 (17.99)
  GGT; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  GGT; Week 12; n= 65, 68 | -2.9 (6.68) | -1.9 (18.70)
  GGT; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  GGT; Week 16; n= 65, 68 | -2.1 (10.18) | -1.5 (21.36)
  GGT; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  GGT; Week 20; n= 63, 68 | 1.7 (19.02) | -1.1 (24.50)
  GGT; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  GGT; Week 24; n= 63, 66 | -1.7 (11.83) | -3.3 (22.52)
  GGT; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  GGT; Week 28; n= 62, 66 | -1.9 (11.71) | -3.1 (16.86)
  GGT; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  GGT; Week 32; n= 61, 67 | -1.5 (15.77) | -3.6 (17.87)
  GGT; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  GGT; Week 36; n= 60, 67 | -2.1 (10.64) | -4.7 (14.96)
  GGT; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  GGT; Week 40; n= 61, 66 | -0.2 (16.05) | -0.3 (19.75)
  GGT; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  GGT; Week 44; n= 61, 66 | -2.9 (8.26) | -2.7 (15.25)
  GGT; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  GGT; Week 48; n= 61, 64 | 0.9 (18.91) | -3.0 (16.51)
  GGT; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  GGT; Week 52; n= 60, 65 | -1.6 (16.44) | -4.2 (13.53)
  GGT; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  GGT; Week 56; n= 61, 63 | -5.0 (16.77) | -3.6 (17.02)
  GGT; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  GGT; Week 60; n= 60, 65 | -4.8 (16.45) | -5.6 (15.37)
  Absolute Lactate dehydro; Baseline; n= 68, 68 | 186.5 (47.82) | 179.6 (38.88)
  Lactate dehydro; Week 4; n= 68, 68 | -3.6 (19.73) | -2.3 (27.80)
  Lactate dehydro; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Lactate dehydro; Week 8; n= 67, 66 | -8.2 (29.91) | -5.3 (24.46)
  Lactate dehydro; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Lactate dehydro; Week 12; n= 65, 68 | -2.2 (27.17) | -7.7 (25.56)
  Lactate dehydro; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Lactate dehydro; Week 16; n= 65, 68 | -2.6 (32.13) | -10.6 (26.12)
  Lactate dehydro; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Lactate dehydro; Week 20; n= 63, 68 | 2.2 (26.80) | -13.7 (25.79)
  Lactate dehydro; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Lactate dehydro; Week 24; n= 63, 66 | -4.3 (26.22) | -13.5 (26.99)
  Lactate dehydro; Week 28; n= 61, 66: number analyzed (Participants) | 61 | 66
  Lactate dehydro; Week 28; n= 61, 66 | -8.5 (27.77) | -15.9 (30.44)
  Lactate dehydro; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Lactate dehydro; Week 32; n= 61, 67 | -8.3 (25.49) | -17.1 (24.88)
  Lactate dehydro; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Lactate dehydro; Week 36; n= 60, 67 | -3.6 (36.45) | -16.2 (30.54)
  Lactate dehydro; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Lactate dehydro; Week 40; n= 61, 66 | -4.5 (35.81) | -13.5 (36.31)
  Lactate dehydro; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Lactate dehydro; Week 44; n= 61, 66 | -2.7 (33.40) | -17.0 (31.37)
  Lactate dehydro; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Lactate dehydro; Week 48; n= 61, 64 | 0.8 (43.82) | -19.0 (30.66)
  Lactate dehydro; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Lactate dehydro; Week 52; n= 60, 65 | -0.1 (34.99) | -17.8 (33.45)
  Lactate dehydro; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Lactate dehydro; Week 56; n= 61, 63 | -5.2 (32.69) | -16.0 (30.87)
  Lactate dehydro; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Lactate dehydro; Week 60; n= 60, 65 | -3.5 (34.15) | -12.4 (33.23)

11. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters of Albumin and Protein Levels
Description: Blood samples were collected to evaluate change from Baseline in albumin and protein levels values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
gram per liter (g/L)
  Absolute Albumin; Baseline; n= 68, 68 | 43.4 (2.45) | 43.5 (3.01)
  Albumin; Week 4; n= 68, 68 | -0.6 (2.25) | -0.1 (2.16)
  Albumin; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Albumin; Week 8; n= 67, 66 | -0.8 (2.16) | -0.6 (2.72)
  Albumin; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Albumin; Week 12; n= 65, 68 | -0.2 (2.47) | -0.4 (2.64)
  Albumin; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Albumin; Week 16; n= 65, 68 | -0.6 (2.57) | -0.6 (2.54)
  Albumin; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Albumin; Week 20; n= 63, 68 | -0.1 (2.35) | -0.2 (2.92)
  Albumin; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Albumin; Week 24; n= 63, 66 | 0.0 (2.80) | 0.1 (2.72)
  Albumin; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Albumin; Week 28; n= 62, 66 | -0.2 (2.67) | 0.1 (2.67)
  Albumin; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Albumin; Week 32; n= 61, 67 | -0.4 (2.71) | -0.1 (2.69)
  Albumin; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Albumin; Week 36; n= 60, 67 | -0.1 (2.58) | 0.3 (3.01)
  Albumin; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Albumin; Week 40; n= 61, 66 | -0.2 (2.98) | 0.2 (2.82)
  Albumin; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Albumin; Week 44; n= 61, 66 | 0.3 (2.95) | -0.3 (2.87)
  Albumin; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Albumin; Week 48; n= 61, 64 | -0.4 (2.74) | -0.3 (2.77)
  Albumin; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Albumin; Week 52; n= 60, 65 | -0.5 (2.45) | -0.3 (3.10)
  Albumin; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Albumin; Week 56; n= 61, 63 | -0.7 (2.84) | -0.5 (2.88)
  Albumin; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Albumin; Week 60; n= 60, 65 | -0.9 (2.55) | -0.7 (3.04)
  Absolute Protein; Baseline; n= 68, 68 | 67.7 (4.26) | 67.3 (4.46)
  Protein; Week 4; n= 68, 68 | -0.8 (3.00) | -0.5 (3.19)
  Protein; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Protein; Week 8; n= 67, 66 | -1.5 (2.97) | -0.9 (3.60)
  Protein; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Protein; Week 12; n= 65, 68 | -0.6 (3.57) | -0.6 (3.30)
  Protein; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Protein; Week 16; n= 65, 68 | -0.3 (3.56) | -0.8 (3.93)
  Protein; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Protein; Week 20; n= 63, 68 | 0.0 (3.21) | 0.1 (4.28)
  Protein; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Protein; Week 24; n= 63, 66 | 0.2 (3.99) | 0.0 (3.96)
  Protein; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Protein; Week 28; n= 62, 66 | -0.2 (4.13) | -0.1 (3.59)
  Protein; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Protein; Week 32; n= 61, 67 | -0.5 (4.09) | -0.4 (3.91)
  Protein; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Protein; Week 36; n= 60, 67 | -0.2 (3.82) | 0.2 (4.45)
  Protein; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Protein; Week 40; n= 61, 66 | -0.4 (3.48) | 0.1 (3.98)
  Protein; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Protein; Week 44; n= 61, 66 | 0.4 (4.43) | -0.6 (4.19)
  Protein; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Protein; Week 48; n= 61, 64 | -0.5 (3.94) | -0.5 (4.29)
  Protein; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Protein; Week 52; n= 60, 65 | -0.3 (3.75) | -0.4 (4.08)
  Protein; week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Protein; week 56; n= 61, 63 | -0.1 (4.77) | -0.5 (4.21)
  Protein; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Protein; Week 60; n= 60, 65 | -0.4 (5.88) | -0.7 (4.17)

12. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters of Direct, Indirect and Total Bilirubin and Creatinine Levels
Description: Blood samples were collected to evaluate change from Baseline in direct, indirect and total bilirubin and creatinine values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micromole per liter (µmol/L)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
micromole per liter (µmol/L)
  Absolute Total bilirubin; Baseline; n= 68, 68 | 9.8 (6.14) | 8.8 (4.10)
  Total bilirubin; week 4; n= 68, 68 | -0.9 (4.02) | 0.1 (3.48)
  Total bilirubin; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Total bilirubin; Week 8; n= 67, 66 | -1.2 (4.38) | 0.0 (3.50)
  Total bilirubin; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Total bilirubin; Week 12; n= 65, 68 | -0.3 (3.01) | 0.1 (3.27)
  Total bilirubin; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Total bilirubin; Week 16; n= 65, 68 | -1.1 (4.15) | 0.0 (4.14)
  Total bilirubin; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Total bilirubin; Week 20; n= 63, 68 | -0.5 (2.90) | 0.3 (3.57)
  Total bilirubin; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Total bilirubin; Week 24; n= 63, 66 | -0.3 (3.36) | 0.0 (2.71)
  Total bilirubin; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Total bilirubin; Week 28; n= 62, 66 | -0.8 (3.13) | 0.3 (4.43)
  Total bilirubin; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Total bilirubin; Week 32; n= 61, 67 | -1.1 (3.07) | -0.1 (3.63)
  Total bilirubin; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Total bilirubin; Week 36; n= 60, 67 | -0.7 (3.39) | 0.1 (4.09)
  Total bilirubin; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Total bilirubin; Week 40; n= 61, 66 | -0.2 (3.22) | -0.3 (3.78)
  Total bilirubin; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Total bilirubin; Week 44; n= 61, 66 | 0.0 (2.50) | 0.1 (3.64)
  Total bilirubin; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Total bilirubin; Week 48; n= 61, 64 | -0.2 (2.59) | -0.1 (3.77)
  Total bilirubin; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Total bilirubin; Week 52; n= 60, 65 | -0.1 (3.41) | 0.7 (3.92)
  Total bilirubin; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Total bilirubin; Week 56; n= 61, 63 | -0.8 (3.17) | 0.5 (3.24)
  Total bilirubin; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Total bilirubin; Week 60; n= 60, 65 | -0.5 (3.21) | 0.0 (3.42)
  Absolute Creatinine; Baseline; n= 68, 68 | 75.49 (12.878) | 73.00 (12.289)
  Creatinine; Week 4; n= 68, 68 | 0.69 (7.195) | 2.09 (5.533)
  Creatinine; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Creatinine; Week 8; n= 67, 66 | 1.87 (7.505) | 1.15 (6.737)
  Creatinine; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Creatinine; Week 12; n= 65, 68 | 1.50 (9.029) | 0.34 (7.006)
  Creatinine; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Creatinine; Week 16; n= 65, 68 | 1.53 (10.012) | 2.72 (6.702)
  Creatinine; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Creatinine; Week 20; n= 63, 68 | 1.73 (6.916) | 2.60 (7.739)
  Creatinine; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Creatinine; Week 24; n= 63, 66 | 0.74 (7.775) | 0.06 (6.538)
  Creatinine; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Creatinine; Week 28; n= 62, 66 | 0.96 (7.504) | 1.02 (7.764)
  Creatinine; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Creatinine; Week 32; n= 61, 67 | 1.89 (9.809) | 1.85 (8.589)
  Creatinine; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Creatinine; Week 36; n= 60, 67 | 1.42 (6.957) | 0.40 (7.839)
  Creatinine; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Creatinine; Week 40; n= 61, 66 | 1.16 (8.253) | 0.34 (8.119)
  Creatinine; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Creatinine; Week 44; n= 61, 66 | 2.14 (8.991) | 0.04 (9.070)
  Creatinine; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Creatinine; Week 48; n= 61, 64 | 1.53 (7.972) | -2.25 (7.398)
  Creatinine; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Creatinine; Week 52; n= 60, 65 | 0.52 (7.719) | -1.35 (7.182)
  Creatinine; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Creatinine; Week 56; n= 61, 63 | 1.39 (7.367) | -0.30 (8.695)
  Creatinine; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Creatinine; Week 60; n= 60, 65 | 0.34 (7.014) | -1.22 (10.896)
  Absolute Direct bilirubin; Baseline; n= 68, 68 | 2.1 (1.33) | 1.9 (0.98)
  Direct bilirubin; Week 4; n= 68, 68 | 0.0 (1.06) | 0.0 (0.84)
  Direct bilirubin; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Direct bilirubin; Week 8; n= 67, 66 | 0.0 (1.01) | 0.1 (0.96)
  Direct bilirubin; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Direct bilirubin; Week 12; n= 65, 68 | 0.0 (0.97) | 0.0 (1.04)
  Direct bilirubin; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Direct bilirubin; Week 16; n= 65, 68 | -0.2 (0.96) | -0.1 (1.20)
  Direct bilirubin; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Direct bilirubin; Week 20; n= 63, 68 | 0.0 (0.86) | 0.1 (1.03)
  Direct bilirubin; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Direct bilirubin; Week 24; n= 63, 66 | 0.1 (0.90) | 0.0 (0.88)
  Direct bilirubin; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Direct bilirubin; Week 28; n= 62, 66 | -0.1 (1.20) | 0.2 (1.15)
  Direct bilirubin; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Direct bilirubin; Week 32; n= 61, 67 | -0.2 (0.99) | 0.1 (0.99)
  Direct bilirubin; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Direct bilirubin; Week 36; n= 60, 67 | -0.1 (1.11) | 0.1 (1.17)
  Direct bilirubin; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Direct bilirubin; Week 40; n= 61, 66 | 0.0 (1.11) | 0.0 (0.94)
  Direct bilirubin; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Direct bilirubin; Week 44; n= 61, 66 | 0.1 (0.93) | 0.0 (1.12)
  Direct bilirubin; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Direct bilirubin; Week 48; n= 61, 64 | 0.1 (0.99) | 0.0 (1.17)
  Direct bilirubin; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Direct bilirubin; Week 52; n= 60, 65 | 0.1 (1.05) | 0.2 (1.06)
  Direct bilirubin; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Direct bilirubin; Week 56; n= 61, 63 | 0.1 (1.08) | 0.1 (1.06)
  Direct bilirubin; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Direct bilirubin; Week 60; n= 60, 65 | 0.1 (1.10) | 0.1 (1.07)
  Absolute Indirect bilirubin; Baseline; n= 68, 68 | 7.7 (5.09) | 6.9 (3.38)
  Indirect bilirubin; Week 4; n= 68, 68 | -0.8 (3.68) | 0.0 (3.06)
  Indirect bilirubin; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Indirect bilirubin; Week 8; n= 67, 66 | -1.2 (3.86) | -0.1 (2.94)
  Indirect bilirubin; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Indirect bilirubin; Week 12; n= 65, 68 | -0.3 (2.61) | 0.1 (2.79)
  Indirect bilirubin; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Indirect bilirubin; Week 16; n= 65, 68 | -0.9 (3.67) | 0.1 (3.37)
  Indirect bilirubin; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Indirect bilirubin; Week 20; n= 63, 68 | -0.5 (2.37) | 0.2 (3.00)
  Indirect bilirubin; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Indirect bilirubin; Week 24; n= 63, 66 | -0.4 (2.94) | 0.0 (2.37)
  Indirect bilirubin; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Indirect bilirubin; Week 28; n= 62, 66 | -0.7 (2.60) | 0.1 (3.71)
  Indirect bilirubin; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  Indirect bilirubin; Week 32; n= 61, 66 | -0.9 (2.48) | -0.2 (3.02)
  Indirect bilirubin; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Indirect bilirubin; Week 36; n= 60, 67 | -0.6 (2.77) | 0.0 (3.30)
  Indirect bilirubin; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Indirect bilirubin; Week 40; n= 61, 66 | -0.1 (2.56) | -0.2 (3.16)
  Indirect bilirubin; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Indirect bilirubin; Week 44; n= 61, 66 | -0.1 (2.19) | 0.1 (2.99)
  Indirect bilirubin; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Indirect bilirubin; Week 48; n= 61, 64 | -0.3 (2.19) | -0.1 (3.13)
  Indirect bilirubin; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Indirect bilirubin; Week 52; n= 60, 65 | -0.2 (2.84) | 0.5 (3.32)
  Indirect bilirubin; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Indirect bilirubin; Week 56; n= 61, 63 | -0.9 (2.72) | 0.4 (2.64)
  Indirect bilirubin; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Indirect bilirubin; Week 60; n= 60, 65 | -0.6 (2.64) | -0.1 (2.81)

13. Secondary Outcome: Change From Baseline in Calcium, Chloride, Cholesterol, Glucose, High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, Phosphorus, Potassium, Sodium, Urea Nitrogen and Very Low Density Lipoprotein (VLDL) Cholesterol Levels
Description: Blood samples were collected to evaluate change from Baseline in calcium, chloride, cholesterol, glucose, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, phosphorus, potassium, sodium, urea nitrogen and very low density lipoprotein (VLDL) cholesterol values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured. NA indicates that data were not available.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
millimoles per liter (mmol/L)
  Absolute Calcium; Baseline; n= 68, 68 | 2.365 (0.0864) | 2.382 (0.1189)
  Calcium; Week 4; n= 68, 68 | -0.011 (0.0836) | -0.012 (0.1200)
  Calcium; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Calcium; Week 8; n= 67, 66 | -0.013 (0.0877) | -0.010 (0.1003)
  Calcium; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Calcium; Week 12; n= 65, 68 | -0.013 (0.0844) | -0.026 (0.0889)
  Calcium; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Calcium; Week 16; n= 65, 68 | 0.000 (0.1091) | -0.029 (0.1018)
  Calcium; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Calcium; Week 20; n= 63, 68 | 0.002 (0.0882) | -0.016 (0.1032)
  Calcium; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Calcium; Week 24; n= 63, 66 | 0.001 (0.0901) | -0.013 (0.1111)
  Calcium; Week 28; n= 61, 66: number analyzed (Participants) | 61 | 66
  Calcium; Week 28; n= 61, 66 | 0.001 (0.0962) | -0.001 (0.1039)
  Calcium; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Calcium; Week 32; n= 61, 67 | -0.000 (0.0911) | -0.006 (0.0977)
  Calcium; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Calcium; Week 36; n= 60, 67 | -0.006 (0.0931) | -0.006 (0.1133)
  Calcium; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Calcium; Week 40; n= 61, 66 | 0.014 (0.1126) | 0.005 (0.1115)
  Calcium; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Calcium; Week 44; n= 61, 66 | 0.016 (0.1144) | -0.020 (0.1115)
  Calcium; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Calcium; Week 48; n= 61, 64 | -0.007 (0.1007) | -0.018 (0.1002)
  Calcium; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Calcium; Week 52; n= 60, 65 | -0.008 (0.1001) | -0.027 (0.1110)
  Calcium; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Calcium; Week 56; n= 61, 63 | -0.008 (0.0931) | -0.015 (0.0994)
  Calcium; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Calcium; Week 60; n= 60, 65 | -0.025 (0.0946) | -0.019 (0.1058)
  Absolute Chloride; Baseline; n= 68, 68 | 103.4 (2.05) | 104.0 (2.21)
  Chloride; Week 4; n= 68, 68 | 0.6 (1.97) | 0.2 (2.00)
  Chloride; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Chloride; Week 8; n= 67, 66 | 0.9 (2.05) | 0.5 (2.06)
  Chloride; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Chloride; Week 12; n= 65, 68 | 0.7 (2.32) | 0.7 (2.20)
  Chloride; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Chloride; Week 16; n= 65, 68 | 0.5 (2.08) | 0.8 (1.95)
  Chloride; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Chloride; Week 20; n= 63, 68 | 0.3 (2.38) | 0.7 (2.04)
  Chloride; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Chloride; Week 24; n= 63, 66 | 0.6 (2.51) | 0.8 (2.20)
  Chloride; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Chloride; Week 28; n= 62, 66 | 0.7 (2.17) | 0.8 (2.59)
  Chloride; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Chloride; Week 32; n= 61, 67 | 0.4 (2.24) | 0.5 (2.32)
  Chloride; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Chloride; Week 36; n= 60, 67 | 0.8 (2.53) | 0.6 (2.08)
  Chloride; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Chloride; Week 40; n= 61, 66 | 0.9 (2.22) | 0.7 (2.13)
  Chloride; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Chloride; Week 44; n= 61, 66 | 0.5 (2.13) | 0.6 (2.55)
  Chloride; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Chloride; Week 48; n= 61, 64 | 0.5 (2.38) | 0.5 (2.34)
  Chloride; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Chloride; Week 52; n= 60, 65 | 0.3 (2.26) | 0.4 (2.24)
  Chloride; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Chloride; Week 56; n= 61, 63 | 0.7 (2.27) | 0.2 (2.06)
  Chloride; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Chloride; Week 60; n= 60, 65 | 0.4 (2.01) | 0.4 (2.20)
  Absolute Cholesterol; Baseline; n= 68, 68 | 5.771 (1.2033) | 5.788 (1.2386)
  Cholesterol; Week 8; n= 2, 0: number analyzed (Participants) | 2 | 0
  Cholesterol; Week 8; n= 2, 0 | -0.250 (0.1414) |
  Cholesterol; Week 12; n= 1, 0: number analyzed (Participants) | 1 | 0
  Cholesterol; Week 12; n= 1, 0 | 0.050 (NA) — NA indicates that data was not available. |
  Cholesterol; Week 16; n= 1, 1: number analyzed (Participants) | 1 | 1
  Cholesterol; Week 16; n= 1, 1 | -0.400 (NA) — NA indicates that data was not available | -0.300 (NA) — NA indicates that data was not available
  Cholesterol; Week 20; n= 1, 1: number analyzed (Participants) | 1 | 1
  Cholesterol; Week 20; n= 1, 1 | 0.050 (NA) — NA indicates that data was not available | -0.300 (NA) — NA indicates that data was not available
  Cholesterol; Week 24; n= 0, 1: number analyzed (Participants) | 0 | 1
  Cholesterol; Week 24; n= 0, 1 |  | -0.560 (NA) — NA indicates that data was not available
  Cholesterol; Week 36; n= 0, 1: number analyzed (Participants) | 0 | 1
  Cholesterol; Week 36; n= 0, 1 |  | 0.420 (NA) — NA indicates that data was not available
  Cholesterol; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Cholesterol; Week 52; n= 60, 65 | -0.006 (0.9364) | -0.384 (0.8798)
  Cholesterol; Week 56; n= 1, 0: number analyzed (Participants) | 1 | 0
  Cholesterol; Week 56; n= 1, 0 | -0.220 (NA) — NA indicates that data was not available |
  Absolute Glucose; Baseline; n= 68, 68 | 5.76 (2.000) | 5.35 (1.195)
  Glucose; Week 4; n= 68, 68 | 0.27 (1.619) | -0.01 (1.050)
  Glucose; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Glucose; Week 8; n= 67, 66 | 0.09 (1.695) | 0.07 (0.986)
  Glucose; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Glucose; Week 12; n= 65, 68 | 0.27 (1.961) | 0.26 (1.079)
  Glucose; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Glucose; Week 16; n= 65, 68 | 0.03 (1.454) | 0.04 (1.077)
  Glucose; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Glucose; Week 20; n= 63, 68 | 0.25 (1.644) | -0.03 (1.351)
  Glucose; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Glucose; Week 24; n= 63, 66 | 0.02 (1.588) | 0.16 (1.211)
  Glucose; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Glucose; Week 28; n= 62, 66 | 0.14 (1.613) | 0.21 (1.551)
  Glucose; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Glucose; Week 32; n= 61, 67 | -0.03 (1.808) | -0.14 (1.162)
  Glucose; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Glucose; Week 36; n= 60, 67 | 0.11 (1.525) | 0.03 (1.003)
  Glucose; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Glucose; Week 40; n= 61, 66 | 0.34 (1.831) | -0.03 (1.305)
  Glucose; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Glucose; Week 44; n= 61, 66 | 0.21 (1.766) | -0.05 (0.891)
  Glucose; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Glucose; Week 48; n= 61, 64 | 0.32 (2.065) | 0.21 (1.740)
  Glucose; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Glucose; Week 52; n= 60, 65 | -0.17 (1.650) | 0.02 (1.258)
  Glucose; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Glucose; Week 56; n= 61, 63 | 0.01 (1.718) | 0.13 (1.852)
  Glucose; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Glucose; Week 60; n= 60, 65 | 0.20 (1.664) | 0.11 (1.483)
  Absolute HDL cholesterol; Baseline; n= 68, 68 | 1.837 (0.4540) | 1.937 (0.5606)
  HDL cholesterol; Week 8; n= 2, 0: number analyzed (Participants) | 2 | 0
  HDL cholesterol; Week 8; n= 2, 0 | -0.075 (0.0354) |
  HDL cholesterol; Week 12; n= 1, 0: number analyzed (Participants) | 1 | 0
  HDL cholesterol; Week 12; n= 1, 0 | -0.100 (NA) — NA indicates that data was not available |
  HDL cholesterol; Week 16; n= 1, 1: number analyzed (Participants) | 1 | 1
  HDL cholesterol; Week 16; n= 1, 1 | 0.400 (NA) — NA indicates that data was not available | -0.150 (NA) — NA indicates that data was not available
  HDL cholesterol; Week 20; n= 1, 1: number analyzed (Participants) | 1 | 1
  HDL cholesterol; Week 20; n= 1, 1 | 0.000 (NA) — NA indicates that data was not available | -0.250 (NA) — NA indicates that data was not available
  HDL cholesterol; Week 24; n= 0, 1: number analyzed (Participants) | 0 | 1
  HDL cholesterol; Week 24; n= 0, 1 |  | -0.390 (NA) — NA indicates that data was not available.
  HDL cholesterol; Week 36; n= 0, 1: number analyzed (Participants) | 0 | 1
  HDL cholesterol; Week 36; n= 0, 1 |  | 0.400 (NA) — NA indicates that data was not available.
  HDL cholesterol; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  HDL cholesterol; Week 52; n= 60, 65 | -0.045 (0.2832) | -0.150 (0.3146)
  HDL cholesterol; Week 56; n= 1, 0: number analyzed (Participants) | 1 | 0
  HDL cholesterol; Week 56; n= 1, 0 | -0.060 (NA) — NA indicates that data was not available. |
  Absolute LDL cholesterol; Baseline; n= 67, 68: number analyzed (Participants) | 67 | 68
  Absolute LDL cholesterol; Baseline; n= 67, 68 | 3.261 (1.0808) | 3.205 (1.0992)
  LDL cholesterol; Week 8; n= 1, 0: number analyzed (Participants) | 1 | 0
  LDL cholesterol; Week 8; n= 1, 0 | -0.350 (NA) — NA indicates that data was not available. |
  LDL cholesterol; Week 12; n= 1, 0: number analyzed (Participants) | 1 | 0
  LDL cholesterol; Week 12; n= 1, 0 | 0.190 (NA) — NA indicates that data was not available. |
  LDL cholesterol; Week 16; n= 1, 1: number analyzed (Participants) | 1 | 1
  LDL cholesterol; Week 16; n= 1, 1 | -0.730 (NA) — NA indicates that data was not available. | -0.790 (NA) — NA indicates that data was not available.
  LDL cholesterol; Week 20; n= 1, 1: number analyzed (Participants) | 1 | 1
  LDL cholesterol; Week 20; n= 1, 1 | -0.150 (NA) — NA indicates that data was not available. | -0.540 (NA) — NA indicates that data was not available.
  LDL cholesterol; Week 24; n= 0, 1: number analyzed (Participants) | 0 | 1
  LDL cholesterol; Week 24; n= 0, 1 |  | 0.040 (NA) — NA indicates that data was not available.
  LDL cholesterol; Week 36; n= 0, 1: number analyzed (Participants) | 0 | 1
  LDL cholesterol; Week 36; n= 0, 1 |  | 0.250 (NA) — NA indicates that data was not available.
  LDL cholesterol; Week 52; n= 58, 64: number analyzed (Participants) | 58 | 64
  LDL cholesterol; Week 52; n= 58, 64 | 0.016 (0.7717) | -0.215 (0.8079)
  LDL cholesterol; Week 56; n= 1, 0: number analyzed (Participants) | 1 | 0
  LDL cholesterol; Week 56; n= 1, 0 | 0.100 (NA) — NA indicates that data was not available. |
  Absolute Phosphate; Baseline; n= 68, 68 | 1.068 (0.1797) | 1.066 (0.1939)
  Phosphate; Week 4; n= 68, 68 | -0.027 (0.2183) | 0.014 (0.1833)
  Phosphate; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Phosphate; Week 8; n= 67, 66 | -0.004 (0.1577) | 0.024 (0.2239)
  Phosphate; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Phosphate; Week 12; n= 65, 68 | 0.003 (0.1821) | 0.019 (0.2181)
  Phosphate; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Phosphate; Week 16; n= 65, 68 | 0.016 (0.1819) | 0.016 (0.2205)
  Phosphate; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Phosphate; Week 20; n= 63, 68 | -0.001 (0.1611) | 0.019 (0.2087)
  Phosphate; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Phosphate; Week 24; n= 63, 66 | -0.042 (0.1565) | 0.007 (0.2142)
  Phosphate; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Phosphate; Week 28; n= 62, 66 | -0.025 (0.1819) | 0.003 (0.2539)
  Phosphate; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Phosphate; Week 32; n= 61, 67 | -0.018 (0.1975) | 0.040 (0.2172)
  Phosphate; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Phosphate; Week 36; n= 60, 67 | -0.038 (0.2159) | 0.023 (0.2260)
  Phosphate; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Phosphate; Week 40; n= 61, 66 | -0.029 (0.1822) | 0.026 (0.2213)
  Phosphate; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Phosphate; Week 44; n= 61, 66 | -0.018 (0.2104) | 0.041 (0.2240)
  Phosphate; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Phosphate; Week 48; n= 61, 64 | -0.053 (0.1931) | -0.020 (0.2443)
  Phosphate; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Phosphate; Week 52; n= 60, 65 | 0.005 (0.1939) | 0.053 (0.2988)
  Phosphate; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Phosphate; Week 56; n= 61, 63 | 0.019 (0.2962) | 0.043 (0.3066)
  Phosphate; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Phosphate; Week 60; n= 60, 65 | -0.035 (0.2125) | -0.007 (0.2322)
  Absolute Potassium; Baseline; n= 68, 68 | 4.11 (0.348) | 4.10 (0.359)
  Potassium; Week 4; n= 68, 68 | 0.05 (0.378) | -0.02 (0.345)
  Potassium; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Potassium; Week 8; n= 67, 66 | 0.01 (0.309) | 0.02 (0.323)
  Potassium; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Potassium; Week 12; n= 65, 68 | -0.04 (0.318) | 0.01 (0.296)
  Potassium; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Potassium; Week 16; n= 65, 68 | 0.06 (0.340) | 0.05 (0.317)
  Potassium; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Potassium; Week 20; n= 63, 68 | 0.08 (0.382) | 0.01 (0.372)
  Potassium; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Potassium; Week 24; n= 63, 66 | -0.02 (0.298) | 0.04 (0.350)
  Potassium; Week 28; n= 61, 66: number analyzed (Participants) | 61 | 66
  Potassium; Week 28; n= 61, 66 | 0.07 (0.338) | 0.10 (0.382)
  Potassium; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Potassium; Week 32; n= 61, 67 | 0.04 (0.340) | 0.11 (0.305)
  Potassium; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Potassium; Week 36; n= 60, 67 | 0.02 (0.291) | 0.01 (0.351)
  Potassium; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Potassium; Week 40; n= 61, 66 | 0.08 (0.419) | 0.14 (0.313)
  Potassium; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Potassium; Week 44; n= 61, 66 | 0.08 (0.383) | 0.09 (0.341)
  Potassium; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Potassium; Week 48; n= 61, 64 | 0.09 (0.367) | 0.05 (0.349)
  Potassium; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Potassium; Week 52; n= 60, 65 | 0.05 (0.344) | 0.01 (0.329)
  Potassium; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Potassium; Week 56; n= 61, 63 | 0.08 (0.379) | 0.08 (0.378)
  Potassium; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Potassium; Week 60; n= 60, 65 | 0.00 (0.358) | 0.10 (0.390)
  Absolute Sodium; Baseline; n= 68, 68 | 139.8 (2.03) | 140.3 (1.83)
  Sodium; Week 4; n= 68, 68 | 0.2 (1.86) | 0.3 (2.03)
  Sodium; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Sodium; Week 8; n= 67, 66 | 0.4 (2.06) | 0.2 (1.89)
  Sodium; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Sodium; Week 12; n= 65, 68 | 0.1 (1.99) | -0.1 (2.28)
  Sodium; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Sodium; Week 16; n= 65, 68 | 0.0 (1.46) | -0.1 (1.91)
  Sodium; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Sodium; Week 20; n= 63, 68 | 0.0 (1.88) | 0.1 (2.09)
  Sodium; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Sodium; Week 24; n= 63, 66 | 0.2 (1.94) | 0.0 (1.95)
  Sodium; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Sodium; Week 28; n= 62, 66 | 0.5 (1.71) | 0.0 (2.23)
  Sodium; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Sodium; Week 32; n= 61, 67 | 0.3 (1.92) | 0.1 (2.13)
  Sodium; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Sodium; Week 36; n= 60, 67 | 0.4 (2.10) | 0.0 (1.95)
  Sodium; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Sodium; Week 40; n= 61, 66 | 0.2 (2.42) | 0.0 (2.18)
  Sodium; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Sodium; Week 44; n= 61, 66 | 0.1 (1.77) | -0.2 (2.02)
  Sodium; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Sodium; Week 48; n= 61, 64 | 0.1 (2.03) | -0.4 (1.97)
  Sodium; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Sodium; Week 52; n= 60, 65 | 0.4 (1.79) | -0.2 (2.17)
  Sodium; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Sodium; Week 56; n= 61, 63 | 0.4 (2.15) | -0.5 (2.08)
  Sodium; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Sodium; Week 60; n= 60, 65 | -0.1 (2.04) | -0.3 (2.36)
  Absolute Urea; Baseline; n= 68, 68 | 5.94 (1.451) | 5.79 (1.629)
  Urea; Week 4; n= 68, 68 | -0.08 (1.412) | 0.09 (1.241)
  Urea; Week 8; n= 67, 66: number analyzed (Participants) | 67 | 66
  Urea; Week 8; n= 67, 66 | -0.23 (1.564) | 0.20 (1.206)
  Urea; Week 12; n= 65, 68: number analyzed (Participants) | 65 | 68
  Urea; Week 12; n= 65, 68 | -0.15 (1.414) | -0.10 (1.217)
  Urea; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Urea; Week 16; n= 65, 68 | -0.07 (1.569) | 0.00 (1.317)
  Urea; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Urea; Week 20; n= 63, 68 | -0.21 (1.465) | -0.23 (1.286)
  Urea; Week 24; n= 63, 66: number analyzed (Participants) | 63 | 66
  Urea; Week 24; n= 63, 66 | -0.28 (1.513) | -0.12 (1.172)
  Urea; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Urea; Week 28; n= 62, 66 | -0.21 (1.525) | -0.22 (1.350)
  Urea; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Urea; Week 32; n= 61, 67 | -0.11 (1.320) | -0.23 (1.359)
  Urea; Week 36; n= 60, 67: number analyzed (Participants) | 60 | 67
  Urea; Week 36; n= 60, 67 | -0.27 (1.407) | -0.32 (1.391)
  Urea; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Urea; Week 40; n= 61, 66 | -0.44 (1.377) | -0.23 (1.375)
  Urea; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Urea; Week 44; n= 61, 66 | -0.32 (1.731) | -0.19 (1.698)
  Urea; Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Urea; Week 48; n= 61, 64 | -0.36 (1.422) | -0.09 (1.429)
  Urea; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Urea; Week 52; n= 60, 65 | -0.19 (1.737) | -0.18 (1.128)
  Urea; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Urea; Week 56; n= 61, 63 | -0.11 (1.495) | -0.13 (1.539)
  Urea; Week 60; n= 60, 65: number analyzed (Participants) | 60 | 65
  Urea; Week 60; n= 60, 65 | -0.09 (1.546) | -0.10 (1.170)
  Absolute VLDL cholesterol; Baseline; n= 67, 68: number analyzed (Participants) | 67 | 68
  Absolute VLDL cholesterol; Baseline; n= 67, 68 | 0.680 (0.2846) | 0.646 (0.2841)
  VLDL cholesterol; Week 8; n= 1, 0: number analyzed (Participants) | 1 | 0
  VLDL cholesterol; Week 8; n= 1, 0 | 0.100 (NA) — NA indicates that data was not available. |
  VLDL cholesterol; Week 12; n= 1, 0: number analyzed (Participants) | 1 | 0
  VLDL cholesterol; Week 12; n= 1, 0 | -0.040 (NA) — NA indicates that data was not available. |
  VLDL cholesterol; Week 16; n= 1, 1: number analyzed (Participants) | 1 | 1
  VLDL cholesterol; Week 16; n= 1, 1 | -0.070 (NA) — NA indicates that data was not available. | 0.640 (NA) — NA indicates that data was not available.
  VLDL cholesterol; Week 20; n= 1, 1: number analyzed (Participants) | 1 | 1
  VLDL cholesterol; Week 20; n= 1, 1 | 0.200 (NA) — NA indicates that data was not available. | 0.490 (NA) — NA indicates that data was not available.
  VLDL cholesterol; Week 24; n= 0, 1: number analyzed (Participants) | 0 | 1
  VLDL cholesterol; Week 24; n= 0, 1 |  | -0.210 (NA) — NA indicates that data was not available.
  VLDL cholesterol; Week 36; n= 0, 1: number analyzed (Participants) | 0 | 1
  VLDL cholesterol; Week 36; n= 0, 1 |  | -0.230 (NA) — NA indicates that data was not available.
  VLDL cholesterol; Week 52; n= 58, 64: number analyzed (Participants) | 58 | 64
  VLDL cholesterol; Week 52; n= 58, 64 | -0.019 (0.3229) | -0.051 (0.1927)
  VLDL cholesterol; Week 56; n= 1, 0: number analyzed (Participants) | 1 | 0
  VLDL cholesterol; Week 56; n= 1, 0 | -0.260 (NA) — NA indicates that data was not available. |

14. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Troponin Levels
Description: Blood samples were collected to evaluate change from Baseline in troponin values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
µg/L
  Absolute Troponin; Baseline; n= 68, 68 | 0.013 (0.0110) | 0.013 (0.0092)
  Troponin; Week 4; n= 68, 66: number analyzed (Participants) | 68 | 66
  Troponin; Week 4; n= 68, 66 | -0.001 (0.0106) | 0.008 (0.0717)
  Troponin; Week 8; n= 67, 67: number analyzed (Participants) | 67 | 67
  Troponin; Week 8; n= 67, 67 | -0.002 (0.0111) | 0.001 (0.0089)
  Troponin; Week 12; n= 64, 67: number analyzed (Participants) | 64 | 67
  Troponin; Week 12; n= 64, 67 | -0.002 (0.0108) | -0.001 (0.0053)
  Troponin; Week 16; n= 65, 68: number analyzed (Participants) | 65 | 68
  Troponin; Week 16; n= 65, 68 | -0.002 (0.0104) | 0.002 (0.0272)
  Troponin; Week 20; n= 61, 68: number analyzed (Participants) | 61 | 68
  Troponin; Week 20; n= 61, 68 | -0.002 (0.0105) | -0.001 (0.0089)
  Troponin; Week 24; n= 62, 67: number analyzed (Participants) | 62 | 67
  Troponin; Week 24; n= 62, 67 | -0.002 (0.0098) | 0.004 (0.0535)
  Troponin; Week 28; n= 63, 66: number analyzed (Participants) | 63 | 66
  Troponin; Week 28; n= 63, 66 | -0.003 (0.0102) | -0.002 (0.0090)
  Troponin; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Troponin; Week 32; n= 61, 67 | -0.003 (0.0100) | -0.002 (0.0092)
  Troponin; Week 36; n= 61, 67: number analyzed (Participants) | 61 | 67
  Troponin; Week 36; n= 61, 67 | -0.002 (0.0107) | 0.000 (0.0185)
  Troponin; Week 40; n= 61, 66: number analyzed (Participants) | 61 | 66
  Troponin; Week 40; n= 61, 66 | -0.001 (0.0117) | -0.002 (0.0090)
  Troponin; Week 44; n= 61, 65: number analyzed (Participants) | 61 | 65
  Troponin; Week 44; n= 61, 65 | -0.000 (0.0068) | -0.001 (0.0095)
  Troponin; Week 48; n= 60, 65: number analyzed (Participants) | 60 | 65
  Troponin; Week 48; n= 60, 65 | 0.017 (0.1479) | -0.001 (0.0101)
  Troponin; Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Troponin; Week 52; n= 60, 65 | -0.002 (0.0114) | -0.001 (0.0111)
  Troponin; Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Troponin; Week 56; n= 61, 63 | -0.003 (0.0112) | -0.002 (0.0086)
  Troponin; Week 60; n= 59, 65: number analyzed (Participants) | 59 | 65
  Troponin; Week 60; n= 59, 65 | -0.003 (0.0109) | -0.001 (0.0093)

15. Secondary Outcome: Change From Baseline in Hematology Parameters of Basophils, Eosinophil, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets Levels
Description: Blood samples were collected to evaluate change from Baseline in basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelet values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
10^9 cells/L
  Absolute Basophils; Baselin; n= 68, 68 | 0.030 (0.0253) | 0.028 (0.0236)
  Basophils; Week 4; n= 66, 66: number analyzed (Participants) | 66 | 66
  Basophils; Week 4; n= 66, 66 | -0.002 (0.0302) | -0.007 (0.0282)
  Basophils; Week 8; n= 65, 66: number analyzed (Participants) | 65 | 66
  Basophils; Week 8; n= 65, 66 | 0.005 (0.0285) | -0.002 (0.0261)
  Basophils; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Basophils; Week 12; n= 63, 65 | 0.007 (0.0351) | -0.007 (0.0222)
  Basophils; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Basophils; Week 16; n= 64, 68 | 0.005 (0.0333) | -0.004 (0.0295)
  Basophils; Week 20; n= 61, 66: number analyzed (Participants) | 61 | 66
  Basophils; Week 20; n= 61, 66 | 0.005 (0.0338) | -0.002 (0.0287)
  Basophils; Week 24; n= 61, 66: number analyzed (Participants) | 61 | 66
  Basophils; Week 24; n= 61, 66 | 0.004 (0.0341) | -0.002 (0.0328)
  Basophils; Week 28; n= 62, 65: number analyzed (Participants) | 62 | 65
  Basophils; Week 28; n= 62, 65 | 0.006 (0.0411) | -0.005 (0.0297)
  Basophils; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  Basophils; Week 32; n= 61, 66 | 0.010 (0.0467) | 0.002 (0.0355)
  Basophils; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Basophils; Week 36; n= 60, 66 | 0.009 (0.0321) | 0.005 (0.0424)
  Basophils; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Basophils; Week 40; n= 61, 65 | 0.005 (0.0357) | -0.002 (0.0356)
  Basophils; Week 44; n= 59, 61: number analyzed (Participants) | 59 | 61
  Basophils; Week 44; n= 59, 61 | 0.008 (0.0328) | 0.000 (0.0296)
  Basophils; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Basophils; Week 48; n= 59, 64 | 0.003 (0.0408) | -0.004 (0.0300)
  Basophils; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Basophils; Week 52; n= 60, 64 | 0.004 (0.0289) | -0.003 (0.0284)
  Basophils; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Basophils; Week 56; n= 59, 61 | 0.009 (0.0381) | -0.003 (0.0286)
  Basophils; Week 60; n= 58, 64: number analyzed (Participants) | 58 | 64
  Basophils; Week 60; n= 58, 64 | 0.002 (0.0316) | -0.006 (0.0248)
  Absolute Eosinophils; Baseline; n= 68, 68 | 0.362 (0.5835) | 0.398 (0.8415)
  Eosinophils; Week 4; n= 66, 66: number analyzed (Participants) | 66 | 66
  Eosinophils; Week 4; n= 66, 66 | -0.054 (0.3309) | -0.339 (0.6794)
  Eosinophils; Week 8; n= 65, 66: number analyzed (Participants) | 65 | 66
  Eosinophils; Week 8; n= 65, 66 | 0.103 (0.2921) | -0.370 (0.8092)
  Eosinophils; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Eosinophils; Week 12; n= 63, 65 | 0.027 (0.3515) | -0.364 (0.8407)
  Eosinophils; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Eosinophils; Week 16; n= 64, 68 | 0.058 (0.4092) | -0.355 (0.8280)
  Eosinophils; Week 20; n= 61, 66: number analyzed (Participants) | 61 | 66
  Eosinophils; Week 20; n= 61, 66 | 0.162 (0.5900) | -0.347 (0.8266)
  Eosinophils; Week 24; n= 61, 66: number analyzed (Participants) | 61 | 66
  Eosinophils; Week 24; n= 61, 66 | 0.136 (0.4044) | -0.364 (0.8211)
  Eosinophils; Week 28; n= 62, 65: number analyzed (Participants) | 62 | 65
  Eosinophils; Week 28; n= 62, 65 | 0.172 (0.4365) | -0.360 (0.8258)
  Eosinophils; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  Eosinophils; Week 32; n= 61, 66 | 0.079 (0.3759) | -0.347 (0.8310)
  Eosinophils; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Eosinophils; Week 36; n= 60, 66 | 0.086 (0.3758) | -0.347 (0.8388)
  Eosinophils; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Eosinophils; Week 40; n= 61, 65 | 0.022 (0.4448) | -0.358 (0.8396)
  Eosinophils; Week 44; n= 59, 61: number analyzed (Participants) | 59 | 61
  Eosinophils; Week 44; n= 59, 61 | 0.051 (0.4472) | -0.365 (0.8604)
  Eosinophils; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Eosinophils; Week 48; n= 59, 64 | 0.109 (0.3873) | -0.364 (0.8540)
  Eosinophils; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Eosinophils; Week 52; n= 60, 64 | 0.055 (0.3764) | -0.341 (0.8456)
  Eosinophils; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Eosinophils; Week 56; n= 59, 61 | 0.071 (0.4137) | -0.351 (0.8624)
  Eosinophils; Week 60; n= 58, 64: number analyzed (Participants) | 58 | 64
  Eosinophils; Week 60; n= 58, 64 | 0.111 (0.4666) | -0.302 (0.8352)
  Absolute Leukocytes; Baseline; n= 68, 68 | 9.91 (2.714) | 9.54 (3.130)
  Leukocytes; Week 4; 66, 66: number analyzed (Participants) | 66 | 66
  Leukocytes; Week 4; 66, 66 | -0.11 (2.109) | -0.77 (2.356)
  Leukocytes; Week 8; n= 65, 66: number analyzed (Participants) | 65 | 66
  Leukocytes; Week 8; n= 65, 66 | -0.18 (2.562) | -0.83 (2.511)
  Leukocytes; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Leukocytes; Week 12; n= 63, 65 | -0.53 (1.765) | -1.24 (2.716)
  Leukocytes; ; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Leukocytes; ; Week 16; n= 64, 68 | 0.01 (2.567) | -1.16 (2.827)
  Leukocytes; Week 20; n= 61, 66: number analyzed (Participants) | 61 | 66
  Leukocytes; Week 20; n= 61, 66 | -0.13 (2.269) | -1.43 (2.649)
  Leukocytes; Week 24; n= 61, 66: number analyzed (Participants) | 61 | 66
  Leukocytes; Week 24; n= 61, 66 | -0.73 (2.110) | -1.47 (2.738)
  Leukocytes; Week 28; n= 62, 65: number analyzed (Participants) | 62 | 65
  Leukocytes; Week 28; n= 62, 65 | -0.01 (2.297) | -1.66 (2.804)
  Leukocytes; week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  Leukocytes; week 32; n= 61, 66 | -0.33 (2.218) | -1.54 (2.725)
  Leukocytes; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Leukocytes; Week 36; n= 60, 66 | -0.17 (2.501) | -1.37 (2.578)
  Leukocytes; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Leukocytes; Week 40; n= 61, 65 | 0.17 (2.912) | -1.28 (3.284)
  Leukocytes; Week 44; n= 59, 61: number analyzed (Participants) | 59 | 61
  Leukocytes; Week 44; n= 59, 61 | 0.25 (3.166) | -1.57 (2.198)
  Leukocytes; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Leukocytes; Week 48; n= 59, 64 | -0.10 (3.092) | -1.46 (2.546)
  Leukocytes; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Leukocytes; Week 52; n= 60, 64 | -0.12 (3.114) | -1.50 (2.521)
  Leukocytes; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Leukocytes; Week 56; n= 59, 61 | -0.05 (3.357) | -1.50 (2.840)
  Leukocytes; Week 60; n= 58, 64: number analyzed (Participants) | 58 | 64
  Leukocytes; Week 60; n= 58, 64 | 0.19 (3.533) | -1.20 (2.396)
  Absolute Lymphocytes; Baseline; n= 68, 68 | 1.638 (0.9375) | 1.508 (0.8230)
  Lymphocytes; Week 4; n= 66, 66: number analyzed (Participants) | 66 | 66
  Lymphocytes; Week 4; n= 66, 66 | 0.031 (0.8990) | 0.145 (0.7485)
  Lymphocytes; Week 8; n= 65, 66: number analyzed (Participants) | 65 | 66
  Lymphocytes; Week 8; n= 65, 66 | 0.245 (0.8804) | -0.048 (0.6388)
  Lymphocytes; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Lymphocytes; Week 12; n= 63, 65 | 0.160 (0.9043) | -0.071 (0.7665)
  Lymphocytes; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Lymphocytes; Week 16; n= 64, 68 | 0.078 (1.0337) | 0.079 (0.7254)
  Lymphocytes; Week 20; n= 61, 66: number analyzed (Participants) | 61 | 66
  Lymphocytes; Week 20; n= 61, 66 | 0.137 (0.7984) | 0.127 (0.7096)
  Lymphocytes; Week 24; n= 61, 66: number analyzed (Participants) | 61 | 66
  Lymphocytes; Week 24; n= 61, 66 | 0.056 (0.8778) | 0.011 (0.8077)
  Lymphocytes; Week 28; n= 62, 65: number analyzed (Participants) | 62 | 65
  Lymphocytes; Week 28; n= 62, 65 | 0.261 (1.0966) | 0.004 (0.7328)
  Lymphocytes; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  Lymphocytes; Week 32; n= 61, 66 | 0.244 (0.9633) | 0.031 (0.7986)
  Lymphocytes; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Lymphocytes; Week 36; n= 60, 66 | 0.156 (1.0399) | 0.031 (0.5939)
  Lymphocytes; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Lymphocytes; Week 40; n= 61, 65 | 0.064 (1.0537) | 0.037 (0.6391)
  Lymphocytes; Week 44; n= 59, 61: number analyzed (Participants) | 59 | 61
  Lymphocytes; Week 44; n= 59, 61 | 0.130 (0.8773) | 0.059 (0.6471)
  Lymphocytes; Week 48; n=59, 64: number analyzed (Participants) | 59 | 64
  Lymphocytes; Week 48; n=59, 64 | 0.106 (0.8396) | 0.035 (0.7368)
  Lymphocytes; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Lymphocytes; Week 52; n= 60, 64 | 0.144 (0.9262) | 0.031 (0.6244)
  Lymphocytes; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Lymphocytes; Week 56; n= 59, 61 | 0.200 (0.8356) | 0.128 (0.7824)
  Lymphocytes; Week 60; n= 58, 64: number analyzed (Participants) | 58 | 64
  Lymphocytes; Week 60; n= 58, 64 | 0.076 (0.8821) | -0.101 (0.6848)
  Absolute Monocytes; Baseline; n= 68, 68 | 0.377 (0.2126) | 0.405 (0.2376)
  Monocytes; week 4; n= 66, 66: number analyzed (Participants) | 66 | 66
  Monocytes; week 4; n= 66, 66 | 0.038 (0.2444) | 0.014 (0.2127)
  Monocytes; Week 8; n= 65, 66: number analyzed (Participants) | 65 | 66
  Monocytes; Week 8; n= 65, 66 | 0.052 (0.2271) | 0.039 (0.1988)
  Monocytes; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Monocytes; Week 12; n= 63, 65 | 0.077 (0.2468) | -0.004 (0.1985)
  Monocytes; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Monocytes; Week 16; n= 64, 68 | 0.086 (0.2790) | 0.031 (0.2157)
  Monocytes; Week 20; n= 61, 66: number analyzed (Participants) | 61 | 66
  Monocytes; Week 20; n= 61, 66 | 0.132 (0.2684) | 0.030 (0.1967)
  Monocytes; Week 24; n= 61, 66: number analyzed (Participants) | 61 | 66
  Monocytes; Week 24; n= 61, 66 | 0.061 (0.2290) | 0.013 (0.2412)
  Monocytes; Week 28; n= 62, 65: number analyzed (Participants) | 62 | 65
  Monocytes; Week 28; n= 62, 65 | 0.107 (0.2363) | 0.035 (0.2350)
  Monocytes; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  Monocytes; Week 32; n= 61, 66 | 0.108 (0.2839) | 0.057 (0.2069)
  Monocytes; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Monocytes; Week 36; n= 60, 66 | 0.089 (0.2992) | 0.072 (0.2416)
  Monocytes; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Monocytes; Week 40; n= 61, 65 | 0.084 (0.2495) | 0.050 (0.2096)
  Monocytes; Week 44; n= 59, 61: number analyzed (Participants) | 59 | 61
  Monocytes; Week 44; n= 59, 61 | 0.090 (0.2494) | 0.077 (0.2176)
  Monocytes; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Monocytes; Week 48; n= 59, 64 | 0.078 (0.2261) | 0.025 (0.2235)
  Monocytes; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Monocytes; Week 52; n= 60, 64 | 0.075 (0.2407) | 0.024 (0.2098)
  Monocytes; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Monocytes; Week 56; n= 59, 61 | 0.051 (0.2104) | 0.037 (0.2303)
  Monocytes; Week 60; n= 58, 64: number analyzed (Participants) | 58 | 64
  Monocytes; Week 60; n= 58, 64 | 0.052 (0.2600) | 0.001 (0.2165)
  Absolute Neutrophils; Baseline; n= 68, 68 | 7.500 (2.7424) | 7.198 (2.9732)
  Neutrophils; Week 4; n= 66, 66: number analyzed (Participants) | 66 | 66
  Neutrophils; Week 4; n= 66, 66 | -0.124 (2.6170) | -0.583 (2.2703)
  Neutrophils; Week 8; n= 65, 66: number analyzed (Participants) | 65 | 66
  Neutrophils; Week 8; n= 65, 66 | -0.572 (2.6791) | -0.443 (2.56476)
  Neutrophils; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Neutrophils; Week 12; n= 63, 65 | -0.797 (2.2948) | -0.799 (2.6278)
  Neutrophils; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Neutrophils; Week 16; n= 64, 68 | -0.222 (2.7666) | -0.914 (2.6034)
  Neutrophils; Week 20; n= 61, 66: number analyzed (Participants) | 61 | 66
  Neutrophils; Week 20; n= 61, 66 | -0.560 (2.3679) | -1.243 (2.6857)
  Neutrophils; Week 24; n= 61, 66: number analyzed (Participants) | 61 | 66
  Neutrophils; Week 24; n= 61, 66 | -0.980 (2.3151) | -1.120 (2.8349)
  Neutrophils; Week 28; n= 62, 65: number analyzed (Participants) | 62 | 65
  Neutrophils; Week 28; n= 62, 65 | -0.555 (2.3719) | -1.335 (2.9428)
  Neutrophils; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  Neutrophils; Week 32; n= 61, 66 | -0.762 (2.4952) | -1.286 (2.6995)
  Neutrophils; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Neutrophils; Week 36; n= 60, 66 | -0.509 (2.8231) | -1.131 (2.4261)
  Neutrophils; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Neutrophils; Week 40; n= 61, 65 | -0.009 (3.0467) | -1.010 (3.3999)
  Neutrophils; Week 44; n= 59, 61: number analyzed (Participants) | 59 | 61
  Neutrophils; Week 44; n= 59, 61 | -0.020 (3.3497) | -1.344 (2.1031)
  Neutrophils; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Neutrophils; Week 48; n= 59, 64 | -0.403 (3.2656) | -1.151 (2.5806)
  Neutrophils; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Neutrophils; Week 52; n= 60, 64 | -0.391 (3.4463) | -1.211 (2.2815)
  Neutrophils; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Neutrophils; Week 56; n= 59, 61 | -0.381 (3.4297) | -1.311 (3.0024)
  Neutrophils; Week 60; n= 58, 64: number analyzed (Participants) | 58 | 64
  Neutrophils; Week 60; n= 58, 64 | -0.048 (3.5724) | -0.795 (2.6501)
  Absolute Platelets; Baseline; n= 68, 68 | 259.8 (61.16) | 270.3 (60.86)
  Platelets; Week 4; n= 66, 67: number analyzed (Participants) | 66 | 67
  Platelets; Week 4; n= 66, 67 | 4.5 (38.14) | -1.4 (33.79)
  Platelets; Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  Platelets; Week 8; n= 66, 66 | 5.0 (43.97) | 4.1 (26.48)
  Platelets; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Platelets; Week 12; n= 63, 65 | 3.1 (50.60) | -4.3 (37.89)
  Platelets; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Platelets; Week 16; n= 64, 68 | 15.4 (71.20) | 1.8 (40.25)
  Platelets; Week 20; n= 61, 68: number analyzed (Participants) | 61 | 68
  Platelets; Week 20; n= 61, 68 | 12.3 (49.92) | 6.1 (52.76)
  Platelets; Week 24; n= 62, 65: number analyzed (Participants) | 62 | 65
  Platelets; Week 24; n= 62, 65 | 10.9 (50.38) | -4.2 (40.07)
  Platelets; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Platelets; Week 28; n= 62, 66 | 13.3 (55.12) | 5.4 (41.57)
  Platelets; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Platelets; Week 32; n= 61, 67 | 12.1 (45.36) | 0.7 (43.85)
  Platelets; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Platelets; Week 36; n= 60, 66 | 9.3 (42.64) | 0.6 (37.87)
  Platelets; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Platelets; Week 40; n= 61, 65 | 14.7 (45.63) | 2.0 (42.12)
  Platelets; Week 44; n= 60, 63: number analyzed (Participants) | 60 | 63
  Platelets; Week 44; n= 60, 63 | 19.3 (48.88) | 4.9 (40.27)
  Platelets; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Platelets; Week 48; n= 59, 64 | 14.2 (53.93) | 5.4 (44.80)
  Platelets; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Platelets; Week 52; n= 60, 64 | 14.7 (48.19) | -3.7 (46.34)
  Platelets; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Platelets; Week 56; n= 59, 61 | 20.3 (47.35) | -1.0 (48.51)
  Platelets; Week 60; n= 59, 64: number analyzed (Participants) | 59 | 64
  Platelets; Week 60; n= 59, 64 | 13.0 (50.07) | -2.0 (41.32)

16. Secondary Outcome: Change From Baseline in Hematology Parameters of Mean Corpuscle Hemoglobin Concentration (MCHC) and Hemoglobin Levels
Description: Blood samples were collected to evaluate change from Baseline in MCHC and hemoglobin values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
g/L
  Absolute MCHC; Baseline; n= 68, 68 | 324.9 (7.53) | 324.4 (7.37)
  MCHC; Week 4; n= 66, 67: number analyzed (Participants) | 66 | 67
  MCHC; Week 4; n= 66, 67 | -1.2 (6.02) | -1.1 (5.92)
  MCHC; Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  MCHC; Week 8; n= 66, 66 | -1.5 (6.69) | -1.5 (6.86)
  MCHC; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  MCHC; Week 12; n= 63, 65 | -1.3 (7.73) | 0.3 (6.60)
  MCHC; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  MCHC; Week 16; n= 64, 68 | -2.3 (7.11) | -2.1 (7.88)
  MCHC; Week 20; n= 61, 68: number analyzed (Participants) | 61 | 68
  MCHC; Week 20; n= 61, 68 | -2.2 (6.65) | -1.2 (7.88)
  MCHC; Week 24; n= 62, 66: number analyzed (Participants) | 62 | 66
  MCHC; Week 24; n= 62, 66 | -3.2 (10.19) | -2.6 (7.39)
  MCHC; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  MCHC; Week 28; n= 62, 66 | -4.3 (7.07) | -2.6 (7.33)
  MCHC; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  MCHC; Week 32; n= 61, 67 | -6.6 (8.19) | -3.6 (7.56)
  MCHC; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  MCHC; Week 36; n= 60, 66 | -4.7 (8.05) | -3.3 (8.37)
  MCHC; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  MCHC; Week 40; n= 61, 65 | -4.5 (8.04) | -3.2 (8.96)
  MCHC; Week 44; n= 60, 64: number analyzed (Participants) | 60 | 64
  MCHC; Week 44; n= 60, 64 | -4.7 (8.51) | -4.5 (9.40)
  MCHC; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  MCHC; Week 48; n= 59, 64 | -6.0 (8.03) | -4.8 (10.56)
  MCHC; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  MCHC; Week 52; n= 60, 64 | -5.2 (7.79) | -5.3 (7.72)
  MCHC; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  MCHC; Week 56; n= 59, 61 | -6.9 (7.74) | -5.3 (7.47)
  MCHC; Week 60; n= 59, 64: number analyzed (Participants) | 59 | 64
  MCHC; Week 60; n= 59, 64 | -7.5 (7.41) | -4.7 (9.90)
  Absolute Hemoglobin; Baseline; n= 68, 68 | 141.6 (12.67) | 140.6 (12.99)
  Hemoglobin; Week 4; n= 66, 67: number analyzed (Participants) | 66 | 67
  Hemoglobin; Week 4; n= 66, 67 | -2.3 (6.86) | -1.8 (6.43)
  Hemoglobin; Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  Hemoglobin; Week 8; n= 66, 66 | -2.5 (7.56) | -1.1 (6.28)
  Hemoglobin; Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Hemoglobin; Week 12; n= 63, 65 | -1.6 (8.28) | -2.2 (7.17)
  Hemoglobin; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Hemoglobin; Week 16; n= 64, 68 | -1.6 (8.24) | -1.9 (7.64)
  Hemoglobin; Week 20; n= 61, 68: number analyzed (Participants) | 61 | 68
  Hemoglobin; Week 20; n= 61, 68 | -0.3 (6.85) | -1.4 (7.64)
  Hemoglobin; Week 24; n= 62, 66: number analyzed (Participants) | 62 | 66
  Hemoglobin; Week 24; n= 62, 66 | -1.1 (8.06) | -1.6 (8.51)
  Hemoglobin; Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Hemoglobin; Week 28; n= 62, 66 | -1.3 (7.48) | -1.3 (8.94)
  Hemoglobin; Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Hemoglobin; Week 32; n= 61, 67 | -1.3 (8.03) | -1.6 (9.22)
  Hemoglobin; Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Hemoglobin; Week 36; n= 60, 66 | -0.2 (8.50) | -0.4 (10.23)
  Hemoglobin; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Hemoglobin; Week 40; n= 61, 65 | 0.1 (8.35) | -0.9 (9.74)
  Hemoglobin; Week 44; n= 60, 64: number analyzed (Participants) | 60 | 64
  Hemoglobin; Week 44; n= 60, 64 | 0.7 (9.59) | -1.9 (10.47)
  Hemoglobin; Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Hemoglobin; Week 48; n= 59, 64 | 0.5 (8.20) | -1.9 (11.07)
  Hemoglobin; Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Hemoglobin; Week 52; n= 60, 64 | 0.1 (8.57) | -1.9 (10.36)
  Hemoglobin; Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Hemoglobin; Week 56; n= 59, 61 | -1.5 (9.92) | -1.9 (11.48)
  Hemoglobin; Week 60; n= 59, 64: number analyzed (Participants) | 59 | 64
  Hemoglobin; Week 60; n= 59, 64 | -1.8 (9.86) | -2.4 (11.36)

17. Secondary Outcome: Change From Baseline in Hematology Parameters of Mean Corpuscle Volume (MCV) Levels
Description: Blood samples were collected to evaluate change from Baseline in MCV values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
femtoliter (fL)
  Absolute, Baseline; n= 68, 68 | 94.8 (9.02) | 94.8 (6.14)
  Week 4; n= 66, 67: number analyzed (Participants) | 66 | 67
  Week 4; n= 66, 67 | 0.4 (1.67) | 0.0 (2.33)
  Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  Week 8; n= 66, 66 | 0.3 (2.50) | 0.0 (2.58)
  Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Week 12; n= 63, 65 | 0.2 (2.00) | -0.7 (2.30)
  Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Week 16; n= 64, 68 | 0.0 (2.22) | -0.4 (2.94)
  Week 20; n= 61, 68: number analyzed (Participants) | 61 | 68
  Week 20; n= 61, 68 | -0.3 (1.87) | -0.9 (2.66)
  Week 24; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 24; n= 62, 66 | -0.5 (2.21) | -1.0 (2.92)
  Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 28; n= 62, 66 | -0.4 (2.86) | -1.4 (3.48)
  Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Week 32; n= 61, 67 | -0.2 (3.01) | -1.7 (3.56)
  Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Week 36; n= 60, 66 | -0.5 (3.55) | -1.9 (3.74)
  Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Week 40; n= 61, 65 | -0.9 (4.09) | -1.4 (3.73)
  Week 44; n= 60, 64: number analyzed (Participants) | 60 | 64
  Week 44; n= 60, 64 | -1.2 (5.06) | -1.5 (3.91)
  Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Week 48; n= 59, 64 | -1.1 (5.96) | -1.5 (4.04)
  Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Week 52; n= 60, 64 | -0.8 (6.52) | -1.3 (4.29)
  Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Week 56; n= 59, 61 | -0.5 (6.47) | -1.0 (4.15)
  Week 60; n= 59, 64: number analyzed (Participants) | 59 | 64
  Week 60; n= 59, 64 | -0.6 (6.57) | -1.0 (4.49)

18. Secondary Outcome: Change From Baseline in Hematology Parameters of Mean Corpuscle Hemoglobin (MCH) Levels
Description: Blood samples were collected to evaluate change from Baseline in MCH values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Picogram (pg)
  Absolute, Baseline; n= 68, 68 | 30.77 (2.902) | 30.77 (2.255)
  Week 4; n= 66, 67: number analyzed (Participants) | 66 | 67
  Week 4; n= 66, 67 | 0.04 (0.331) | -0.12 (0.785)
  Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  Week 8; n= 66, 66 | -0.02 (0.950) | -0.16 (0.653)
  Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Week 12; n= 63, 65 | -0.04 (0.550) | -0.17 (0.769)
  Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Week 16; n= 64, 68 | -0.21 (0.845) | -0.34 (0.769)
  Week 20; n= 61, 68: number analyzed (Participants) | 61 | 68
  Week 20; n= 61, 68 | -0.28 (0.665) | -0.41 (0.851)
  Week 24; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 24; n= 62, 66 | -0.45 (1.270) | -0.59 (0.959)
  Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 28; n= 62, 66 | -0.51 (0.618) | -0.70 (1.184)
  Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Week 32; n= 61, 67 | -0.66 (0.764) | -0.88 (1.368)
  Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Week 36; n= 60, 66 | -0.60 (0.910) | -0.90 (1.395)
  Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Week 40; n= 61, 65 | -0.67 (1.171) | -0.79 (1.390)
  Week 44; n= 60, 64: number analyzed (Participants) | 60 | 64
  Week 44; n= 60, 64 | -0.78 (1.566) | -0.95 (1.484)
  Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Week 48; n= 59, 64 | -0.87 (1.745) | -0.96 (1.654)
  Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Week 52; n= 60, 64 | -0.69 (1.908) | -0.95 (1.585)
  Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Week 56; n= 59, 61 | -0.79 (2.056) | -0.83 (1.713)
  Week 60; n= 59, 64: number analyzed (Participants) | 59 | 64
  Week 60; n= 59, 64 | -0.86 (2.094) | -0.80 (1.818)

19. Secondary Outcome: Change From Baseline in Hematology Parameters of Erythrocytes Levels
Description: Blood samples were collected to evaluate change from Baseline in erythrocytes values at Baseline throughout the 52 weeks study treatment and 8-weeks follow up period. Baseline values were taken at Visit 2 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
10^12 cells/L
  Absolute, Baseline; n= 68, 68 | 4.64 (0.511) | 4.58 (0.456)
  Week 4; n= 66, 67: number analyzed (Participants) | 66 | 67
  Week 4; n= 66, 67 | -0.07 (0.228) | -0.03 (0.226)
  Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  Week 8; n= 66, 66 | -0.07 (0.278) | -0.01 (0.211)
  Week 12; n= 63, 65: number analyzed (Participants) | 63 | 65
  Week 12; n= 63, 65 | -0.04 (0.273) | -0.04 (0.252)
  Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Week 16; n= 64, 68 | -0.02 (0.266) | -0.01 (0.243)
  Week 20; n= 61, 68: number analyzed (Participants) | 61 | 68
  Week 20; n= 61, 68 | 0.03 (0.243) | 0.03 (0.252)
  Week 24; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 24; n= 62, 66 | 0.02 (0.252) | 0.05 (0.265)
  Week 28; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 28; n= 62, 66 | 0.03 (0.286) | 0.08 (0.264)
  Week 32; n= 61, 67: number analyzed (Participants) | 61 | 67
  Week 32; n= 61, 67 | 0.06 (0.300) | 0.09 (0.273)
  Week 36; n= 60, 66: number analyzed (Participants) | 60 | 66
  Week 36; n= 60, 66 | 0.08 (0.314) | 0.14 (0.299)
  Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  Week 40; n= 61, 65 | 0.09 (0.274) | 0.09 (0.270)
  Week 44; n= 60, 64: number analyzed (Participants) | 60 | 64
  Week 44; n= 60, 64 | 0.13 (0.332) | 0.08 (0.260)
  Week 48; n= 59, 64: number analyzed (Participants) | 59 | 64
  Week 48; n= 59, 64 | 0.14 (0.293) | 0.10 (0.271)
  Week 52; n= 60, 64: number analyzed (Participants) | 60 | 64
  Week 52; n= 60, 64 | 0.10 (0.309) | 0.09 (0.251)
  Week 56; n= 59, 61: number analyzed (Participants) | 59 | 61
  Week 56; n= 59, 61 | 0.06 (0.365) | 0.07 (0.284)
  Week 60; n= 59, 64: number analyzed (Participants) | 59 | 64
  Week 60; n= 59, 64 | 0.07 (0.384) | 0.05 (0.318)

20. Secondary Outcome: Number of Participants With Anti-Mepolizumab Antibodies
Description: Blood samples were collected for the determination of anti-Mepolizumab antibodies. Participants who showed presence of anti-Mepolizumab antibody were termed as 'positive' and those who did not have anti-Mepolizumab antibody in blood sample were termed as 'negative'. Participants who did not have a positive ADA assay prior to the first dose of investigational product were included in the analysis.
Time Frame: Up to Week 60
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 67 | 66
Participants
  Negative | 66 | 65
  Positive | 1 | 1

21. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Levels
Description: SBP and DBP were measured from Baseline throughout follow-up (till Week 60) before injection with the participant sitting, having rested in this position for at least 5 minutes before reading. The Baseline value was taken at Visit 2 and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mm of Hg)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
millimeter of mercury (mm of Hg)
  Absolute SBP; Baseline; n= 68, 68 | 127.46 (17.794) | 122.46 (14.134)
  SBP; Week 4; n= 68, 68 | 0.47 (15.865) | 0.93 (12.370)
  SBP; Week 8; n= 67, 68: number analyzed (Participants) | 67 | 68
  SBP; Week 8; n= 67, 68 | 0.07 (14.192) | 1.29 (11.066)
  SBP; Week 12; n= 66, 68: number analyzed (Participants) | 66 | 68
  SBP; Week 12; n= 66, 68 | -1.12 (14.380) | -1.41 (12.071)
  SBP; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  SBP; Week 16; n= 64, 68 | -0.97 (16.630) | -0.41 (11.579)
  SBP; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  SBP; Week 20; n= 63, 68 | -0.97 (15.028) | -0.85 (12.019)
  SBP; Week 24; n= 63, 67: number analyzed (Participants) | 63 | 67
  SBP; Week 24; n= 63, 67 | -1.54 (15.449) | -1.57 (12.824)
  SBP; Week 28; n= 63, 67: number analyzed (Participants) | 63 | 67
  SBP; Week 28; n= 63, 67 | -0.06 (14.337) | -0.15 (13.240)
  SBP; Week 32; n= 62, 67: number analyzed (Participants) | 62 | 67
  SBP; Week 32; n= 62, 67 | -2.35 (14.027) | 0.04 (11.181)
  SBP; Week 36; n= 62, 67: number analyzed (Participants) | 62 | 67
  SBP; Week 36; n= 62, 67 | 1.02 (14.663) | 0.48 (14.397)
  SBP; Week 40; n= 62, 66: number analyzed (Participants) | 62 | 66
  SBP; Week 40; n= 62, 66 | 0.90 (14.202) | 1.27 (12.075)
  SBP; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  SBP; Week 44; n= 61, 66 | 1.41 (16.143) | -0.36 (13.694)
  SBP; Week 48; n= 61, 65: number analyzed (Participants) | 61 | 65
  SBP; Week 48; n= 61, 65 | -0.41 (17.140) | -0.22 (12.351)
  SBP: Week 52; n= 61, 65: number analyzed (Participants) | 61 | 65
  SBP: Week 52; n= 61, 65 | -1.03 (13.200) | -0.32 (13.091)
  SBP; Week 56; n= 62, 63: number analyzed (Participants) | 62 | 63
  SBP; Week 56; n= 62, 63 | 0.06 (15.216) | 1.02 (13.559)
  SBP; Week 60; n= 61, 65: number analyzed (Participants) | 61 | 65
  SBP; Week 60; n= 61, 65 | 0.61 (15.627) | -0.63 (11.656)
  Absolute DBP; Baseline; n= 68, 68 | 80.21 (10.127) | 76.22 (9.646)
  DBP; Week 4; n= 68, 68 | -2.26 (10.046) | 1.01 (10.130)
  DBP; Week 8; n= 67, 68: number analyzed (Participants) | 67 | 68
  DBP; Week 8; n= 67, 68 | -2.04 (8.461) | -0.34 (10.078)
  DBP; Week 12; n= 66, 68: number analyzed (Participants) | 66 | 68
  DBP; Week 12; n= 66, 68 | -1.92 (10.115) | -0.37 (9.167)
  DBP; Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  DBP; Week 16; n= 64, 68 | -1.36 (10.237) | 0.46 (9.824)
  DBP; Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  DBP; Week 20; n= 63, 68 | -1.25 (8.092) | -1.19 (9.214)
  DBP; Week 24; n= 63, 67: number analyzed (Participants) | 63 | 67
  DBP; Week 24; n= 63, 67 | -2.24 (8.751) | -1.16 (9.629)
  DBP; Week 28; n= 63, 67: number analyzed (Participants) | 63 | 67
  DBP; Week 28; n= 63, 67 | -2.02 (9.939) | 0.36 (10.071)
  DBP; Week 32; n= 62, 67: number analyzed (Participants) | 62 | 67
  DBP; Week 32; n= 62, 67 | -4.27 (9.313) | -0.49 (10.652)
  DBP; Week 36; n= 62, 67: number analyzed (Participants) | 62 | 67
  DBP; Week 36; n= 62, 67 | -1.97 (10.995) | 0.16 (10.988)
  DBP; Week 40; n= 62, 66: number analyzed (Participants) | 62 | 66
  DBP; Week 40; n= 62, 66 | -0.48 (9.625) | -0.03 (8.868)
  DBP; Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  DBP; Week 44; n= 61, 66 | -0.79 (9.930) | -1.03 (9.595)
  DBP; Week 48; n= 61, 65: number analyzed (Participants) | 61 | 65
  DBP; Week 48; n= 61, 65 | -3.26 (10.466) | -1.71 (9.239)
  DBP; Week 52; n= 61, 65: number analyzed (Participants) | 61 | 65
  DBP; Week 52; n= 61, 65 | -3.66 (10.628) | -0.06 (9.236)
  DBP; Week 56; n= 62, 63: number analyzed (Participants) | 62 | 63
  DBP; Week 56; n= 62, 63 | -3.48 (10.570) | 0.11 (8.899)
  DBP; Week 60; n= 61, 65 | -2.54 (11.278) | -0.45 (9.836)

22. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured from Baseline throughout follow-up (till Week 60) before injection with the participant sitting, having rested in this position for at least 5 minutes before reading. The Baseline value was taken at Visit 2 and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
beats per minute (bpm)
  Absolute Baseline; n= 68, 68 | 77.38 (13.763) | 75.75 (10.404)
  Week 4; n= 68, 68 | 2.01 (12.294) | 1.87 (10.543)
  Week 8; n= 67, 68: number analyzed (Participants) | 67 | 68
  Week 8; n= 67, 68 | 0.97 (10.718) | -1.01 (10.304)
  Week 12; n= 66, 68: number analyzed (Participants) | 66 | 68
  Week 12; n= 66, 68 | 1.52 (12.393) | -0.12 (10.855)
  Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Week 16; n= 64, 68 | 0.59 (11.287) | 0.44 (11.411)
  Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Week 20; n= 63, 68 | 1.03 (11.521) | -0.56 (9.687)
  Week 24; n= 63, 67: number analyzed (Participants) | 63 | 67
  Week 24; n= 63, 67 | 0.79 (12.134) | 0.37 (10.057)
  Week 28; n= 62, 67: number analyzed (Participants) | 62 | 67
  Week 28; n= 62, 67 | 1.29 (10.439) | 0.16 (10.093)
  Week 32; n= 62, 67: number analyzed (Participants) | 62 | 67
  Week 32; n= 62, 67 | 1.60 (11.703) | -0.31 (10.530)
  Week 36; n= 62, 67: number analyzed (Participants) | 62 | 67
  Week 36; n= 62, 67 | 3.47 (12.538) | -0.57 (11.422)
  Week 40; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 40; n= 62, 66 | 2.65 (12.297) | 0.74 (11.669)
  Week 44; n= 61, 66: number analyzed (Participants) | 61 | 66
  Week 44; n= 61, 66 | 3.10 (12.195) | 0.15 (12.763)
  Week 48; n= 61, 65: number analyzed (Participants) | 61 | 65
  Week 48; n= 61, 65 | 3.85 (12.383) | -1.12 (10.315)
  Week 52; n= 61, 65: number analyzed (Participants) | 61 | 65
  Week 52; n= 61, 65 | 1.85 (11.987) | -2.17 (9.596)
  Week 56; n= 62, 63: number analyzed (Participants) | 62 | 63
  Week 56; n= 62, 63 | 2.60 (14.041) | -0.35 (9.986)
  Week 60; n= 61, 65: number analyzed (Participants) | 61 | 65
  Week 60; n= 61, 65 | 1.51 (12.793) | 0.09 (10.280)

23. Secondary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured from Baseline throughout follow-up (till Week 60). The Baseline value was taken at Visit 2 and change from Baseline was defined as post dose visit value minus Baseline value. The analysis was performed on Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
Degree celsius
  Absolute Baseline; n= 68, 68 | 36.52 (0.385) | 36.51 (0.462)
  Week 4; n= 68, 68 | 0.05 (0.439) | -0.04 (0.411)
  Week 8; n= 67,68: number analyzed (Participants) | 67 | 68
  Week 8; n= 67,68 | -0.01 (0.379) | -0.02 (0.425)
  Week 12; n= 66, 68: number analyzed (Participants) | 66 | 68
  Week 12; n= 66, 68 | 0.05 (0.410) | -0.03 (0.447)
  Week 16; n= 64, 68: number analyzed (Participants) | 64 | 68
  Week 16; n= 64, 68 | -0.01 (0.421) | -0.03 (0.432)
  Week 20; n= 63, 68: number analyzed (Participants) | 63 | 68
  Week 20; n= 63, 68 | -0.08 (0.351) | -0.13 (0.376)
  Week 24; n= 62, 67: number analyzed (Participants) | 62 | 67
  Week 24; n= 62, 67 | -0.06 (0.449) | -0.06 (0.389)
  Week 28; n= 63, 67: number analyzed (Participants) | 63 | 67
  Week 28; n= 63, 67 | -0.06 (0.499) | -0.14 (0.411)
  Week 32; n= 62, 67: number analyzed (Participants) | 62 | 67
  Week 32; n= 62, 67 | -0.09 (0.392) | -0.07 (0.355)
  Week 36; n= 62, 67: number analyzed (Participants) | 62 | 67
  Week 36; n= 62, 67 | -0.05 (0.431) | 0.03 (0.468)
  Week 40; n= 62, 66: number analyzed (Participants) | 62 | 66
  Week 40; n= 62, 66 | -0.03 (0.530) | -0.13 (0.406)
  Week 44; n= 61, 65: number analyzed (Participants) | 61 | 65
  Week 44; n= 61, 65 | -0.03 (0.550) | -0.08 (0.396)
  Week 48; n= 61, 64: number analyzed (Participants) | 61 | 64
  Week 48; n= 61, 64 | -0.04 (0.452) | -0.09 (0.414)
  Week 52; n= 60, 65: number analyzed (Participants) | 60 | 65
  Week 52; n= 60, 65 | -0.04 (0.423) | -0.12 (0.541)
  Week 56; n= 61, 63: number analyzed (Participants) | 61 | 63
  Week 56; n= 61, 63 | -0.08 (0.530) | -0.00 (0.402)
  Week 60; n= 61, 64: number analyzed (Participants) | 61 | 64
  Week 60; n= 61, 64 | 0.03 (0.467) | -0.02 (0.479)

24. Secondary Outcome: Mean Change From Baseline in QT Interval Corrected by Fridericia's Method (QTcF) and QT Interval Corrected by Bazett's Method (QTcB) Values
Description: Single measurements of 12-lead electrocardiogram (ECGs) were obtained after 5 minutes rest in a supine position at Baseline throughout the 52 weeks treatment period and 8 weeks follow-up period using an ECG machine. Mean change from Baseline in QTcF and QTcB values were measured. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
milliseconds (msec)
  QTcF; Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  QTcF; Week 8; n= 66, 66 | 0.1 (17.90) | 1.0 (15.03)
  QTcF; Week 16; n= 64, 66: number analyzed (Participants) | 64 | 66
  QTcF; Week 16; n= 64, 66 | 0.8 (15.26) | 0.2 (14.05)
  QTcF; Week 24; n= 60, 66: number analyzed (Participants) | 60 | 66
  QTcF; Week 24; n= 60, 66 | 2.8 (14.43) | 1.9 (16.66)
  QTcF; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  QTcF; Week 32; n= 61, 66 | 6.2 (25.19) | 1.5 (17.16)
  QTcF; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  QTcF; Week 40; n= 61, 65 | -0.5 (15.25) | -0.3 (17.53)
  QTcF; Week 52; n= 58, 64: number analyzed (Participants) | 58 | 64
  QTcF; Week 52; n= 58, 64 | 2.0 (15.96) | 3.0 (16.04)
  QTcF; Week 60; n= 58, 63: number analyzed (Participants) | 58 | 63
  QTcF; Week 60; n= 58, 63 | 3.0 (14.30) | 2.9 (14.97)
  QTcF; Any time post Baseline; n= 68, 68 | 16.9 (23.74) | 15.4 (13.79)
  QTcB; Week 8; n= 66, 66: number analyzed (Participants) | 66 | 66
  QTcB; Week 8; n= 66, 66 | -0.8 (19.05) | 0.9 (17.31)
  QTcB; Week 16; n= 64, 66: number analyzed (Participants) | 64 | 66
  QTcB; Week 16; n= 64, 66 | -0.1 (18.33) | -0.9 (14.76)
  QTcB; Week 24; n= 60, 66: number analyzed (Participants) | 60 | 66
  QTcB; Week 24; n= 60, 66 | 1.4 (17.89) | 1.0 (18.10)
  QTcB; Week 32; n= 61, 66: number analyzed (Participants) | 61 | 66
  QTcB; Week 32; n= 61, 66 | 5.2 (29.63) | 0.0 (19.63)
  QTcB; Week 40; n= 61, 65: number analyzed (Participants) | 61 | 65
  QTcB; Week 40; n= 61, 65 | -0.6 (17.83) | -1.4 (18.88)
  QTcB; Week 52; n= 58, 64: number analyzed (Participants) | 58 | 64
  QTcB; Week 52; n= 58, 64 | 1.8 (17.64) | 0.7 (18.27)
  QTcB; Week 60; n= 58, 63: number analyzed (Participants) | 58 | 63
  QTcB; Week 60; n= 58, 63 | 1.2 (16.56) | 2.7 (17.27)
  QTcB; Any time post Baseline; n= 68, 68 | 18.8 (26.46) | 18.1 (15.28)

25. Secondary Outcome: Maximum Change From Baseline in QTcF and QTcB Values
Description: Single measurements of 12-lead ECGs were obtained after 5 minutes rest in a supine position at Baseline throughout the 52 weeks treatment period and 8 weeks follow-up period using an ECG machine. Maximum change from Baseline in QTcF and QTcB values were measured.
Time Frame: Baseline and up to Week 60
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Mepolizumab 300mg
Number analyzed (Participants) | 68 | 68
msec
  QTcB interval | 18.8 (26.46) | 18.1 (15.28)
  QTcF interval | 16.9 (23.74) | 15.4 (13.79)

ADVERSE EVENTS:
Time Frame: On-treatment Serious Adverse Events (SAEs) and non-serious Adverse Events (AEs) were collected from the start of the study treatment until week 52.
Description: AEs and SAEs were collected in Safety Population which comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo | Mepolizumab 300mg
All-Cause Mortality (participants affected / at risk) | 0/68 | 1/68
Serious Adverse Events (participants affected / at risk) | 18/68 | 12/68
Other Adverse Events (participants affected / at risk) | 61/68 | 65/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | Mepolizumab 300mg (N=68)
Influenza (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Lower respiratory infection (Infections and infestations) | 2 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebellar ischaemia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Pachymeningitis (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Allergic granulomatous angiitis (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | Mepolizumab 300mg (N=68)
Nasopharyngitis (Infections and infestations) | 16 | 12
Sinusitis (Infections and infestations) | 11 | 14
Upper respiratory tract infection (Infections and infestations) | 11 | 14
Bronchitis (Infections and infestations) | 8 | 7
Influenza (Infections and infestations) | 6 | 7
Respiratory tract infection (Infections and infestations) | 8 | 5
Urinary tract infection (Infections and infestations) | 4 | 5
Acute sinusitis (Infections and infestations) | 2 | 6
Conjunctivitis (Infections and infestations) | 4 | 4
Rhinitis (Infections and infestations) | 3 | 5
Ear infection (Infections and infestations) | 6 | 1
Fungal skin infection (Infections and infestations) | 3 | 4
Oral herpes (Infections and infestations) | 3 | 4
Gastroenteritis (Infections and infestations) | 1 | 5
Otitis media (Infections and infestations) | 1 | 3
Viral infection (Infections and infestations) | 1 | 3
Nausea (Gastrointestinal disorders) | 13 | 11
Diarrhoea (Gastrointestinal disorders) | 8 | 12
Vomiting (Gastrointestinal disorders) | 4 | 11
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 10 | 10
Injection site reaction (General disorders) | 7 | 9
Pyrexia (General disorders) | 7 | 7
Asthenia (General disorders) | 3 | 5
Chest pain (General disorders) | 5 | 1
Injection site pain (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 1 | 3
Influenza like illness (General disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Headache (Nervous system disorders) | 12 | 22
Dizziness (Nervous system disorders) | 5 | 3
Paraesthesia (Nervous system disorders) | 3 | 4
Sinus headache (Nervous system disorders) | 3 | 2
Migraine (Nervous system disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3
Vision blurred (Eye disorders) | 2 | 4
Cataract (Eye disorders) | 2 | 3
Eye pruritus (Eye disorders) | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 2 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 5
Ear discomfort (Ear and labyrinth disorders) | 4 | 1
Alanine aminotransferase increased (Investigations) | 0 | 5
Weight increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 3
Insomnia (Psychiatric disorders) | 4 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 3
Hot flush (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.